CLINICAL TRIAL: NCT03056157
Title: Psychosocial Rehabilitation After Moral Injury and Loss With Adaptive Disclosure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); San Diego Veterans Healthcare System (U.S. Federal Agency); Central Texas Veterans Health Care System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2135-I; RX-15-005 (Other Grant/Funding Number: Office of Research and Development)
Record Dates: First submitted 2017-01-31; First posted 2017-02-17 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Post-traumatic Stress Disorder; Moral Injury; Traumatic Loss
Keywords: Moral Injury; Post-traumatic Stress Disorder; Traumatic Loss; Adaptive Disclosure; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adaptive Disclosure for Moral Injury and Loss (Experimental): AD-MIL is a manualized, 12-session individual psychotherapy designed to improve functioning and to reduce PTSD symptoms by facilitating Veterans doing corrective things in their life to heal and repair traumatic loss and moral injuries. The change agents are: (1) emotional-processing of traumatic loss and moral injuries and motivating a healing and action plan by writing therapeutic letters (e.g., to a lost unit member, to victims of personal transgressions, to people who transgressed); (2) skills training and behavioral contracting to improve functioning and targeting moral injury- and traumatic loss-related psychological and behavioral obstacles to positive and potentially habilitative engagements in occupational, relationship, and family roles; and (3) teaching self- and other-compassion and mindfulness. The goal is to redress the functional impact of moral emotions (anger, shame).
  Interventions: Behavioral: Adaptive Disclosure for Moral Injury and Loss
- Present Centered Therapy (Active Comparator): PCT is a manualized evidenced-based PTSD treatment used in several large-scale PTSD trials that focuses on improving day-to-day functioning. It incorporates the essential therapeutic elements common to different types of psychotherapies, including supportive empathic listening and unconditional positive regard. The therapist plays an active role but does not impart any systematic training. The focus is to create an understanding of how the symptoms of PTSD are related to day-to-day difficulties and to help patients develop new, more adaptive functional responses to these stressors with a problem-focused and problem-solving approach. In prior trials, PCT showed equivalent change to active therapies at the last follow-up. The VA offers PCT as an evidence-based therapy for PTSD.
  Interventions: Behavioral: Present Centered Therapy

INTERVENTIONS:
Behavioral: Adaptive Disclosure for Moral Injury and Loss — AD-MIL is a manualized, 12-session individual psychotherapy designed to improve functioning and to reduce PTSD symptoms by facilitating Veterans doing corrective things in their life to heal and repair traumatic loss and moral injuries. The change agents are: (1) emotional-processing of traumatic loss and moral injuries and motivating a healing and action plan by writing therapeutic letters (e.g., to a lost unit member, to victims of personal transgressions, to people who transgressed); (2) skills training and behavioral contracting to improve functioning and targeting moral injury- and traumatic loss-related psychological and behavioral obstacles to positive and potentially habilitative engagements in occupational, relationship, and family roles; and (3) teaching self- and other-compassion and mindfulness. The goal is to redress the functional impact of moral emotions (anger, shame).
  Other Names: AD-MIL
  Arms: Adaptive Disclosure for Moral Injury and Loss
Behavioral: Present Centered Therapy — Participants randomized to the PCT arm will receive 12 sessions of therapy focused on day-to-day functional problems with no focus on trauma or re-visiting past experiences
  Other Names: PCT
  Arms: Present Centered Therapy

SUMMARY:
The aim of this study was to determine the efficacy of Adaptive Disclosure for Moral Injury and Loss (AD-MIL), a combat-specific psychotherapy for war-related PTSD stemming from Moral Injury (MI) and traumatic loss (TL) with Iraq and Afghanistan War Veterans with PTSD. AD-MIL will be compared to Present Centered Therapy (PCT). AD-MIL is a modified version of Adaptive Disclosure (AD), which has been modified and extended to solely treat MI and TL by targeting psychological and behavioral obstacles to occupational, relationship, and family functioning, as well as quality of life. PCT is a manualized evidenced-based PTSD treatment used to address functioning problems in several large-scale PTSD trials. The primary end-point was psychosocial functioning (improvements in social, educational and occupational functions). Secondary end-points included PTSD, depression, moral emotions (anger, shame, and guilt), alcohol use, self-compassion, and mindful/valued living.

DETAILED DESCRIPTION:
The investigators conducted a multi-site randomized trial comparing Adaptive Disclosure for Moral Injury and Loss (AD-MIL; an expanded version of Adaptive Disclosure) for war-related PTSD stemming from Moral Injury (MI) and traumatic loss (TL) to Present Centered Therapy (PCT; Frost et al., 2014). The primary endpoint was psychosocial functioning. The investigators had six hypotheses:

A: Functional and behavioral changes:

A.1. Immediately post-treatment, and 3- and 6-months post-treatment, Veterans with PTSD randomized to AD-MIL will have greater reductions in social, educational, and occupational disability.

A.2. COVID-19 aim. In the extended time period for the trial, at the post-treatment, or post-treatment and 3-months post-treatment intervals (depending on when the participant was randomized), Veterans with PTSD randomized to AD-MIL will have greater reductions in social, educational and occupational disability (the investigators also explored whether there would be greater PTSD and depression symptom reduction in this interval).

B: Mental health changes:

B.3. AD-MIL will lead to greater reductions in PTSD symptom severity and a smaller percentage of PTSD cases.

B.4. AD-MIL will lead to greater reductions in depressive symptoms. B.5. AD-MIL will lead to greater reductions in shame and guilt B.6. AD-MIL will lead to greater reductions in psychological distress.

Exploratory hypotheses: AD-MIL will lead to greater reductions in aggressive behaviors, suicidal ideation, and alcohol use, and greater increases in compassion for the self and others and social connectedness.

BACKGROUND PTSD is a functionally disabling condition among war Veterans. Approximately 20% of Veterans of post-9-11 operations have clinically significant PTSD and suffer from a variety of co-morbid mental and physical health conditions. They also have extensive functional impairments, aggressive and risky behaviors, and reduced quality of life. Although considerable gains have been made in the VA's dissemination of PTSD treatments that are highly effective with civilian trauma, these therapies have been shown to work considerably less well for war trauma. The investigators have argued that this is partly due to a lack of attention to the military culture and warrior ethos and the unique harms of war trauma, namely, moral injury (MI) and traumatic loss (TL). In addition, PTSD treatments have failed to demonstrate an impact on functioning and quality of life, problems that are no less impacted by the warzone trauma. Instead, symptom change is typically the sole metric of success, and functional deficits are rarely considered. The investigators argue that PTSD symptoms should be conceptualized and targeted as part of the fabric of the whole Veteran and his or her context. The investigators aimed to fill a care-gap in the VA by creating an evidence-based treatment for war-related PTSD stemming from MI and TL, focusing on improving psychosocial functioning. The investigators extended Adaptive Disclosure to treat MI and TL (AD-MIL) by: (1) facilitating emotional-processing of TL and MIs and a healing and action plan by letter writing tasks to the lost person or, depending on the nature of the MI, the person or persons harmed by transgressive acts (MI stemming from personal actions or the failure to act) or the person or persons who were the transgressors (MI stemming from being the victim of others' transgressions or bearing witness to grave transgressive acts); (2) skills training and behavioral contracting to improve functioning and targeting MI- and TL-related psychological and behavioral obstacles to habilitative engagements in occupational, relationship, and family roles; and (3) teaching self- and other-compassion and mindfulness. If found to be effective, AD-MIL will fill a care-gap in the VA, reduce PTSD patients' suffering, and help Veterans reclaim or establish positive relationships, work roles, and self-care routines.

METHOD Overview: The VA sites were Boston, Minneapolis, San Francisco, San Diego, and Central Texas. The coordinating/lead site was VA Boston led by the study PI, Brett Litz, PhD. The trial followed the consensus recommendations for clinical trials in the VA (VA ORD, 2008): (1) clearly defined target symptoms: functional and clinical outcomes were operationalized; (2) reliable and valid measures: assessment tools were selected for their content relevance and psychometric properties; (3) use of blind evaluators of outcome: the evaluator was independent and blind to treatment condition. This assessor reminded participants to help maintain their blind; (4) assessor training: the independent evaluator was carefully trained to criteria and monitored on an ongoing basis; (5) manualized, replicable, specific treatment programs; (6) there was unbiased assignment to treatment arms and (7) treatment adherence: sessions were be recorded, and a random percentage was used to assess treatment integrity. Adherence to the therapy manuals was monitored by senior supervisors. The investigators followed the CONSORT guidelines for randomization and participant tracking.

Participants: The trial required 148 Veterans (including women and members of diverse ethnic and racial groups) with PTSD as a result of military trauma.

Recruitment: Veterans were recruited and treated at the Minneapolis, San Diego, San Francisco, and Waco VAs. Co-Investigators (Co-Is): (a) provided materials describing the nature of the study and the target populations sought, distributing said materials via formal (e.g., staff meetings) and informal (e.g., bulletin boards) channels; (b) attended clinical staff meetings; (c) gave talks to describe various treatments in staff grand rounds and other contexts (e.g., to trainees); and (d) provided feedback to staff about referred patients.

Assessor Training and Adherence: A co-investigator, Dr. Matt Gray (University of Wyoming) trained the assessors prior to beginning enrollment. Training included reading and viewing training materials, observation of CAPS-5 administration, and supervised administration of at least three CAPS-5s. Dr. Gray has expertise in CAPS-5 training and fidelity monitoring. The assessor was considered trained on CAPS-5 when they matched Dr. Gray on three interviews. To establish matching, Dr. Gray co-rated interviews conducted by the assessor. A match occurred when the assessor and Dr. Gray agreed on the diagnosis and were within 2 severity points on all of the symptom clusters (PTSD criteria B, C, D, and E).

All assessments were audiotaped to ensure that a standardized approach was used across patients (provided that the participant consents). Dr. Gray reviewed a random 10% of the assessments. All recordings were stored on a restricted-access encrypted drive. Selected recordings were transported to Dr. Gray via Federal Express that allows tracking.

Random Assignment: Veterans were assigned to PCT or AD-MIL based on a randomized permuted block scheme, blocked by gender and minority status. Block size for gender and minority status was based on the distribution of these variables at each site. The Boston site used constrained randomization (i.e., biased coin design) if unexpected imbalance arose in gender and minority distribution across treatment groups.

Treatment Fidelity Monitoring: Half-time therapists with Ph.Ds. in clinical or counseling psychology and VA internship experiences treating Veterans with PTSD were trained to deliver AD-MIL and PCT. Training involved a review of the respective manuals and supporting materials, intensive one-on-one training and supervision, and weekly and ad hoc supervision (Dr. Litz for AD-MIL; Dr. Harris for PCT). All sessions were audiotaped. Two random session recordings from a random 20% of the cases were rated to ensure fidelity to each treatment approach.

ANALYSES Data Analysis: The longitudinal and clustered nature of the design produced a multilevel or nested data structure (Raudenbush & Bryk, 2002), with a likelihood of between-subject variability in treatment trajectory over time (e.g., random slopes). In this study, Veterans and therapists were nested (clustered) within performance sites. The lower level (level-1) data consisted of the repeated measures for each individual at each assessment. Level-1 data is nested within upper level (level-2) person-level variables (e.g., study site).

Using SAS 9.4 and R/R Studio, the investigators explored the change trajectory of endpoints over the course of pre-treatment, during-treatment, and post-treatment time intervals. Specifically, the investigators used the linear mixed model regression framework to assess the differential treatment effects of endpoint symptom burden over time. The investigators examined observed measurement scores and specified linear mixed models that best fit the time-change trends (e.g., linear, piecewise). The investigators tested for the presence of random variation, such as between-site cluster effects and between-subject random slopes of treatment effect. The investigators determined the best fit linear mixed effects model as a combination of most appropriate representation of time and empirically-evidenced random and fixed effects.

The linear mixed effects models incorporated clinically relevant time-invariant and time-varying predictors and used Maximum Likelihood Estimation to produce estimates that were unbiased in the presence of random missingness and dropout. These provided an Intent-To-Treat (ITT) analysis that incorporated all available data. Per-protocol and "completer" subset analyses were performed under the same paradigm. Additionally, a subset of subjects who began therapy during the COVID-19 pandemic were identified and analyzed separately; they comprised subjects which began therapy following December 31st, 2020. The tenability of the "At-Random" missingness assumption was assessed and a sensitivity analysis of the results was conducted to determine robustness of the inferences.

Clinical significance: The investigators used a variation of the two-stage Jacobson & Truax (J&T; 1991) method to establish a reasonable cutoff between dysfunctional and functional scores. The investigators first established the cutoff A, defined as the point 2 SDs beyond the range of the pre-therapy mean (cutoff A = M(baseline) - 2 SD(baseline)). Next, the investigators generated a reliable change index (RCI) for each participant to ensure that changes were not due to artifact of measurement error ([x2 - x1]/Sdiff where x1 represents the participant's pre-treatment total score, x2 represents the participant's post-treatment or follow-up total score, and Sdiff is the standard error of difference between the two test scores. Sdiff was calculated from the test-retest reliability of measures. An RCI larger than 1.96 reflects real change. Individuals were classified as recovered (passed both cutoff A and RC criteria), improved (passed RC criterion but not cutoff A), unchanged (passed neither criterion), or deteriorated (passed RC criterion but symptom scores increased) for each follow-up interval. Chi-square analyses were used to compare proportions per arm at each follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Served in an active-duty role within the military since September 2001 (Veterans may be eligible whether or not they were deployed to a warzone)
2. Met the DSM-5 diagnostic criteria for PTSD as a result of military trauma (per Clinician Administered PTSD Scale for DSM-5 [CAPS-5]) and reported non-negligible levels of associated functional impairment (Sheehan Disability Scale [SDS] score = 10)
3. Prospective enrollees must have been willing to commit to 12 consecutive weekly therapy sessions lasting up to 90 minutes in duration and to complete assessment materials.

Exclusion Criteria:

1. Bipolar or psychotic disorders.
2. Current drug or alcohol dependence (other than caffeine or tobacco dependence). Prospective enrollees who had maintained sobriety for at least 6 weeks immediately prior to the time of enrollment may have been eligible.
3. Evidence of traumatic brain injury severe enough to influence the ability to understand and respond to study procedures
4. Suicidal or homicidal ideation severe enough to warrant immediate attention
5. Concurrent enrollment in any treatment that involves: (1) systematic disclosure of troubling trauma-related memories or (2) present-focused psychosocial skills training for PTSD or (3) supportive therapy/case management on a > monthly basis or (4) any individual therapy or (5) newly (< 6 weeks) prescribed pharmacological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett T. Litz, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (5):
- United States (5):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Central Texas Veterans Health Care System Waco VA Medical Center, Waco, TX, Waco, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frost ND, Laska KM, Wampold BE. The evidence for present-centered therapy as a treatment for posttraumatic stress disorder. J Trauma Stress. 2014 Feb;27(1):1-8. doi: 10.1002/jts.21881. PMID 24515534
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Straus MA, Douglas EM. A short form of the Revised Conflict Tactics Scales, and typologies for severity and mutuality. Violence Vict. 2004 Oct;19(5):507-20. doi: 10.1891/vivi.19.5.507.63686. PMID 15844722
- [Background] Weathers FW, Keane TM, Davidson JR. Clinician-administered PTSD scale: a review of the first ten years of research. Depress Anxiety. 2001;13(3):132-56. doi: 10.1002/da.1029. PMID 11387733
- [Background] Batterham PJ, Fairweather-Schmidt AK, Butterworth P, Calear AL, Mackinnon AJ, Christensen H. Temporal effects of separation on suicidal thoughts and behaviours. Soc Sci Med. 2014 Jun;111:58-63. doi: 10.1016/j.socscimed.2014.04.004. Epub 2014 Apr 8. PMID 24768777
- [Background] Forbes D, Hawthorne G, Elliott P, McHugh T, Biddle D, Creamer M, Novaco RW. A concise measure of anger in combat-related posttraumatic stress disorder. J Trauma Stress. 2004 Jun;17(3):249-56. doi: 10.1023/B:JOTS.0000029268.22161.bd. PMID 15253097
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Kubany ES, Haynes SN, Abueg FR, Manke FP, Brennan JM, & Stahura C. Development and validation of the Trauma-Related Guilt Inventory (TRGI). Psychological Assessment. 1996; 8(4): 428-444.
- [Background] Lee RM, Robbins SB. Measuring belongingness: The social connectedness and the social assurance scales. Journal of Counseling Psychology. 1995; 42(2): 232-241.
- [Background] Marx BP. Development & validation of a PTSD-related impairment scale. Boston VA Research Institute.
- [Background] Metalsky GI, Joiner TE. The hopelessness depression symptom questionnaire. Cognitive Therapy and Research. 1997; 21(3): 359-384.
- [Background] Neff KD. The development and validation of a scale to measure self-compassion. Self and identity. 2003; 2(3): 223-250.
- [Background] Øktedalen T, Hagtvet KA, Hoffart A, Langkaas TF, Smucker M. The Trauma Related Shame Inventory: Measuring trauma-related shame among patients with PTSD. Journal of Psychopathology and Behavioral Assessment. 2014; 36(4): 600-615.
- [Background] Raudenbush SW, Bryk AS. Hierarchical linear models: Applications and data analysis methods (Vol 1). Sage; 2002.
- [Background] Sheehan DV. (1983). The Anxiety Disease. New York: Charles Scribner and Sons.
- [Background] Sheehan DV, Harnett-Sheehan K, Raj BA. The measurement of disability. Int Clin Psychopharmacol. 1996 Jun;11 Suppl 3:89-95. doi: 10.1097/00004850-199606003-00015. PMID 8923116
- [Background] Sobell LC, Agrawal S, Sobell MB, Leo GI, Young LJ, Cunningham JA, Simco ER. Comparison of a quick drinking screen with the timeline followback for individuals with alcohol problems. J Stud Alcohol. 2003 Nov;64(6):858-61. doi: 10.15288/jsa.2003.64.858. PMID 14743950
- [Background] Straus MA, Hamby SL, Boney-McCoy SU, Sugarman DB. The revised conflict tactics scales (CTS2) development and preliminary psychometric data. Journal of family issues. 1996; 17(3): 283-316.
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Weathers FW, Litz BT, Keane TM, Palmieri PA, Marx BP, Schnurr PP. The PTSD checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www. ptsd.va.gov. 2013; 10(4): 206.
- [Background] Blais MA, Lenderking WR, Baer L, deLorell A, Peets K, Leahy L, Burns C. Development and initial validation of a brief mental health outcome measure. J Pers Assess. 1999 Dec;73(3):359-73. doi: 10.1207/S15327752JPA7303_5. PMID 10689649
- [Background] Wilson, K. G., Sandoz, E. K., Kitchens, J., & Roberts, M. (2010). The Valued Living Questionnaire: Defining and measuring valued action within a behavioral framework. The Psychological Record, 60(2), 249-272. https://doi.org/10.1007/BF03395706
- [Background] Hwang, J.Y., Plante, T. & Lackey, K. The development of the Santa Clara Brief Compassion Scale: An abbreviation of Sprecher and Fehr's Compassionate Love Scale. Pastoral Psychol 56, 421-428 (2008). https://doi.org/10.1007/s11089-008-0117-2
- [Derived] Litz BT, Yeterian J, Berke D, Lang AJ, Gray MJ, Nienow T, Frankfurt S, Harris JI, Maguen S, Rusowicz-Orazem L. A controlled trial of adaptive disclosure-enhanced to improve functioning and treat posttraumatic stress disorder. J Consult Clin Psychol. 2024 Mar;92(3):150-164. doi: 10.1037/ccp0000873. PMID 38358703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through clinician referral at four VA locations: San Francisco, San Diego, Minneapolis, and Central Texas between January 2018 and November 2021. The first participant was enrolled on January 3rd, 2018 and the last on November 19th, 2021.
Pre-assignment Details: 304 participants were recruited for the study. 96 did not meet inclusion/exclusion criteria, 20 declined to participate, and 14 were excluded for other reasons (e.g., difficult to contact). A total of 174 were randomized.
Groups:
- Present Centered Therapy: Participants randomized to the PCT arm received 12 sessions of therapy focused on improving day-to-day functioning (with no focus on trauma or re-visiting past experiences). PCT is a manualized evidenced-based PTSD treatment used in several large-scale PTSD trials that focuses on improving functioning. It incorporates the essential therapeutic elements common to different types of psychotherapies, including supportive empathic listening and unconditional positive regard. The therapist plays an active role, but does not impart any systematic training. The focus is to create an understanding of how the symptoms of PTSD are related to day-to-day difficulties and to help patients develop new, more adaptive functional responses to these stressors with a problem-focused and problem- solving approach. In prior trials, PCT showed equivalent change to active therapies at the last follow-up. The VA offers PCT as an evidence-based therapy for PTSD.
Period: Overall Study
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Started (Completed baseline assessments.) | 89 | 85
Started Treatment (Attended at Least One Therapy Session) | 80 | 83
Completed Treatment (A participant was considered to have completed treatment if they received twelve sessions within the allotted 16-week interval or were deemed an early completer by their study therapist.) | 59 | 52
Completed 12 Sessions | 56 | 50
Completed 3-month Follow up | 54 | 62
Completed 6-month Follow up | 43 | 41
COVID-19 Cohort (Participants who started the study after December 1, 2020 are considered to be in the COVID-19 cohort.) | 21 | 22
Completed | 59 | 52
Not Completed | 30 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy | Total
Number analyzed (Participants) | 89 | 85 | 174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 85 | 174
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.82 (8.61) | 39.24 (8.61) | 39.02 (8.61)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 69 | 66 | 135
  Gender: Female | 19 | 18 | 37
  Gender: Transgender | 0 | 1 | 1
  Gender: Prefer not to answer | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 21 | 40
  Not Hispanic or Latino | 66 | 58 | 124
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — "Other" is included under "Unknown or Not Recorded" due to table constraints
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 4 | 5 | 9
    Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
    Black or African American | 10 | 9 | 19
    White | 54 | 50 | 104
    More than one race | 5 | 12 | 17
    Unknown or Not Reported | 12 | 7 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 89 | 85 | 174
Sheehan Disability Scale (SDS) [Mean (Standard Deviation); unit: Score on a scale] — The Sheehan Disability Scale (SDS; Sheehan, 1983; Sheehan et al., 1996) is a composite of three self-rated items regarding the degree to which symptoms disrupted work/school, social life, and family life/responsibilities on an 11-point scale ranging from "Not at all" to "Extremely," with an option for "Not applicable". The possible range of scores is 0 to 30. Higher scores indicate greater disability. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 82 | 84 | 166
    (all) | 20.52 (5.14) | 20.43 (5.10) | 20.48 (5.10)
Brief Inventory of Psychosocial Functioning (B-IPF) [Mean (Standard Deviation); unit: Percentage of total possible score] — The Brief Inventory of Psychosocial Functioning (B-IPF; Marx et al., 2013) was used to assess functional gains. It is a 7-item scale indexing overall level of functioning in seven life domains: romantic relationship, relationship with children, family relationships, friendships and socializing, work, training and education, and activities of daily living. Possible scores on the B-IPF range from 0% to 100%, with higher scores indicating more issues in psychosocial functioning. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Percentage of total possible score
    number analyzed (Participants) | 85 | 82 | 167
    (all) | 59.37 (22.14) | 61.06 (19.39) | 60.20 (20.79)
COVID-19 Aim: Sheehan Disability Scale (SDS) [Mean (Standard Deviation); unit: Score on a scale] — The Sheehan Disability Scale (SDS; Sheehan, 1983; Sheehan et al., 1996) is a composite of three self-rated items regarding the degree to which symptoms disrupted work/school, social life, and family life/responsibilities on an 11-point scale ranging from "Not at all" to "Extremely," with an option for "Not applicable". The possible range of scores is 0 to 30. Higher scores indicate greater disability. Population: This analysis is just of participants who started the study after December 1, 2020 (COVID-19 cohort). Additionally, some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 18 | 22 | 40
    (all) | 21.78 (4.52) | 19.82 (5.83) | 20.70 (5.31)
COVID-19 Aim: PTSD Checklist for DSM-5 (PCL-5) [Mean (Standard Deviation); unit: Score on a scale] — The PTSD Checklist for DSM-5 (PCL-5; Weathers et al., 2013) is a 20-item self-report checklist based on the 20 DSM-5 symptoms post-traumatic stress disorder (PTSD). The PCL-5 has been validated as a means of monitoring symptom change during treatment. The 20 items are scored are scored in the past month on a scale from 0 ("not at all") to 4 ("extremely"), generating a total symptom severity score between 0 and 80, with higher scores indicating greater PTSD symptom severity. Population: This analysis is just of participants who started the study after December 1, 2020 (COVID-19 cohort). Additionally, some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 20. | 20 | 40
    (all) | 48.53 (8.84) | 50.62 (11.57) | 49.73 (10.40)
COVID-19 Aim: Clinician-administered PTSD scale for DSM-5 (CAPS-5) [Mean (Standard Deviation); unit: Score on a scale] — The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5; Weathers et al., 2013) is closely modeled on the CAPS-IV, a structured diagnostic interview and gold standard for assessing PTSD. It has excellent psychometric properties and diagnostic efficiency (Weathers, Keane, & Davidson, 2001). The CAPS-5 uses a single 4-point ordinal rating scale to measure symptom severity. These ratings combine information about symptom frequency and intensity obtained by the interviewer. CAPS-5 scores range from 0 to 80, with higher scores indicating greater PTSD symptom severity. Population: This analysis is just of participants who started the study after December 1, 2020 (COVID-19 cohort).
  Score on a scale
    number analyzed (Participants) | 21 | 22 | 43
    (all) | 39.76 (8.89) | 40.86 (9.15) | 40.33 (8.93)
COVID-19 Aim: Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: Score on a scale] — The Patient Health Questionnaire (PHQ-9) is widely used and well-validated measure of symptoms of depression (Kroenke et al., 2001). It scores each of the nine DSM criteria for depression on a scale of 0 ("not at all") to 3 ("nearly every day"). The range of possible scores is 0 to 27. A higher score indicates more frequent depression symptoms. Population: This analysis is just of participants who started the study after December 1, 2020 (COVID-19 cohort). Additionally, some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 17 | 20 | 37
    (all) | 17.31 (5.38) | 14.95 (6.14) | 15.88 (5.88)
PTSD Checklist for DSM-5 (PCL-5) [Mean (Standard Deviation); unit: Score on a scale] — The PTSD Checklist for DSM-5 (PCL-5; Weathers et al., 2013) is a 20-item self-report checklist based on the 20 DSM-5 symptoms post-traumatic stress disorder. The PCL-5 has been validated as a means of monitoring symptom change during treatment. The 20 items are scored are scored in the past month on a scale from "0 = not at all" to "4 = extremely.", generating a total symptom severity score between 0 and 80, with higher scores indicating greater PTSD symptom severity. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 83 | 83 | 166
    (all) | 49.26 (11.43) | 51.66 (10.85) | 50.46 (11.17)
Clinician-administered PTSD scale for DSM-5 (CAPS-5) [Mean (Standard Deviation); unit: Score on a scale] — The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5; Weathers et al., 2013) is closely modeled on the CAPS-IV, a structured diagnostic interview and gold standard for assessing PTSD. It has excellent psychometric properties and diagnostic efficiency (Weathers, Keane, & Davidson, 2001). The CAPS-5 uses a single 4-point ordinal rating scale to measure symptom severity. These ratings combine information about symptom frequency and intensity obtained by the interviewer. CAPS-5 scores range from 0 to 80, with higher scores indicating greater PTSD symptom severity. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale | 36.08 (11.88) | 35.69 (13.60) | 35.89 (12.71)
Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: Score on a scale] — The Patient Health Questionnaire (PHQ-9) is widely used and well-validated measure of symptoms of depression (Kroenke et al., 2001). It scores each of the 9 DSM criteria for depression on a scale of 0 "not at all" to 3 "nearly every day". The range of possible scores is 0 to 27. A higher score indicates more frequent depression symptoms. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 79 | 82 | 161
    (all) | 16.88 (5.43) | 16.62 (5.50) | 16.75 (5.45)
(Lack of) Justification Subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief). [Mean (Standard Deviation); unit: Score on a scale] — The (lack of) Justification subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief; Kubany et al., 1996) is a 4-item measure that assesses guilty thoughts about the justification of one's actions related to a specific traumatic event. Possible scores range from 0 to 4, with higher scores indicating increased guilt. Population: Measure Analysis Population Description: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group
  Score on a scale
    number analyzed (Participants) | 81 | 80 | 161
    (all) | 1.88 (0.98) | 2.00 (0.96) | 1.94 (0.97)
Hindsight-Bias Subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief) [Mean (Standard Deviation); unit: Score on a scale] — The Hindsight-Bias subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief; Kubany et al., 1996) is a 7-item measure that assesses guilty thoughts about the preventability and responsibility of a traumatic event. Possible scores range from 0 to 4, with higher scores indicating increased guilt. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 81 | 80 | 161
    (all) | 1.66 (1.06) | 1.68 (1.04) | 1.67 (1.05)
Wrongdoing Subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief) [Mean (Standard Deviation); unit: Score on a scale] — The Wrongdoing subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief; Kubany et al., 1996) is a 5-item measure that assesses guilty thoughts about wrongdoing tied to a specific traumatic event. Possible scores range from 0 to 4, with higher scores indicating increased guilt. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 84 | 81 | 165
    (all) | 1.71 (1.00) | 1.74 (1.01) | 1.72 (1.00)
Internal Shame Subscale of the Trauma-Related Shame Inventory (TRSI) [Mean (Standard Deviation); unit: Score on a scale] — The Internal Shame Subscale of the Trauma-Related Shame Inventory (TRSI; Øktedalen et al., 2014) is a 12-item self-report instrument designed to assess individuals' negative self-evaluations in the context of their traumatic experiences. Possible scores range from 0 to 36, with higher scores indicating more negative self-evaluations. The measure has demonstrated good construct validity (Øktedalen et al., 2014). Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group
  Score on a scale
    number analyzed (Participants) | 82 | 80 | 162
    (all) | 12.74 (7.94) | 14.23 (9.46) | 13.48 (8.73)
Schwartz Outcome Scale-10 (SOS-10) [Mean (Standard Deviation); unit: Score on a scale] — The Schwartz Outcome Scale-10 (SOS-10; Blais et al., 1999) is a 10-item general mental health outcome measure meant to capture quality of life by assessing psychological health and distress. Possible scores range from 0 to 60 with higher scores indicating better psychological health and lower distress. The SOS-10 has demonstrated good psychometric properties (Blais et al., 1999). Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 85 | 82 | 167
    (all) | 24.94 (9.87) | 25.43 (8.38) | 25.18 (9.14)
Self-Compassion Scale (SCS) [Mean (Standard Deviation); unit: Score on a scale] — The Self Compassion Scale (SCS; Neff, 2003) is a 26-item measure that includes 6 subscales (including Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, and Over-Identification) and measures overall self-compassion. The possible range of scores is 1 to 5, with higher scores indicating higher self-compassion. The SCS has shown good internal consistency reliability as well as good test-retest reliability (Neff, 2003). Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 82 | 81 | 163
    (all) | 2.66 (0.57) | 2.49 (0.56) | 2.58 (0.57)
Dimensions of Anger Reactions (DAR) [Mean (Standard Deviation); unit: Score on a scale] — The Dimensions of Anger Reactions (DAR; Forbes et al., 2004) is a widely used measure of state anger. The measure consists of a 7-item inventory intended to capture anger disposition. Possible scores range from 0 to 56, with higher scores indicating higher state anger. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 85 | 81 | 166
    (all) | 30.27 (12.90) | 32.32 (12.06) | 31.27 (12.50)
Psychological Aggression Subscale of the Revised Conflict Tactics Scale (CTS2) [Mean (Standard Deviation); unit: Score on a scale] — The Psychological Aggression subscale of the Revised Conflict Tactics Scale (CTS2; Straus et al., 1996) was used to measure psychologically aggressive behavior. The subscale consists of 8 items, rated on a scale from 0 ("never") to 6 ("more than 20 times"), with higher scores indicating greater use of aggressive behaviors in the past month. To calculate the annual frequency score, values of 3 through 6 were transformed as follows: 3 = 4, 4 = 8, 5 = 15, 6 = 25. These values were then summed, with higher scores indicating greater frequency. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 85 | 82 | 167
    (all) | 28.94 (31.45) | 26.41 (27.87) | 27.70 (29.68)
Physical Assault Subscale on the Revised Conflict Tactics Scale (CTS2) [Mean (Standard Deviation); unit: Score on a scale] — The physical assault subscale of the Revised Conflict Tactics Scale (CTS2; Straus & Douglas, 2004; Straus et al., 1996) was used to measure occurrence of physically aggressive behavior. The subscale consists of 12 items, rated on a scale from 0 ("never") to 6 ("more than 20 times"), with higher scores indicating greater use of aggressive behaviors in the past month. To calculate the annual frequency score, values of 3 through 6 were transformed as follows: 3 = 4, 4 = 8, 5 = 15, 6 = 25. These values were then summed, with higher scores indicating greater frequency. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 85 | 82 | 167
    (all) | 5.25 (30.27) | 0.96 (3.31) | 3.31 (21.76)
Depressive Symptoms Index - Suicidality Subscale (DSI-SS) [Mean (Standard Deviation); unit: Score on a scale] — The Depressive Symptoms Index - Suicidality Subscale (DSI-SS; Metalsky & Joiner, 1997) is a 4-item scale that focuses on ideation, plans, perceived control over ideation, and impulses for suicide. A review of measures of suicidal ideation and behaviors found that the DSI-SS had excellent internal consistency and concurrent validity (Batterham et al., 2014). Possible scores range from 0 to 12, with higher scores indicating greater severity of suicidal ideation. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 81 | 82 | 163
    (all) | 1.14 (1.62) | 0.93 (1.65) | 1.03 (1.64)
Quick Drinking Screen (QDS) [Mean (Standard Deviation); unit: Drinks per week] — Alcohol abuse was evaluated with the Quick Drinking Screen (QDS; Sobell et al., 2003), a 4-item probe of frequency and quantity of alcohol consumption in the last month. The QDS has very good psychometric characteristics (Sobell et al., 2003). The outcome for this measure used in this study was average drinks per week, calculated by using items 1 and 2 from the screen. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Drinks per week
    number analyzed (Participants) | 85 | 82 | 167
    (all) | 1.92 (3.17) | 1.97 (2.82) | 1.94 (2.99)
Social Connectedness Scale (SCS) [Mean (Standard Deviation); unit: Score on a scale] — The Social Connectedness Scale (SCS; Lee and Robbins, 1995) was used to assess interpersonal closeness. The SCS is an 8-item scale that focuses on individual experiences in a social world (i.e., with peers, friends, and society) and the degree of difficulty in maintaining a sense of closeness. Possible scores range from 8 to 42, with higher scores indicating more social connection. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Score on a scale
    number analyzed (Participants) | 85 | 82 | 167
    (all) | 23.89 (9.69) | 23.57 (8.22) | 23.73 (8.97)
Santa Clara Brief Compassion Scale (SCBSC) [Mean (Standard Deviation); unit: Score on a scale] — The Santa Clara Brief Compassion Scale (SCBSC; Hwang, et al., 2008) is a 5-item short form of the Compassionate Love Scale for Humanity (CLS). Possible scores range from 1 to 7, with higher scores indicating more compassion for humanity. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group
  Score on a scale
    number analyzed (Participants) | 85 | 82 | 167
    (all) | 4.84 (1.76) | 5.00 (1.64) | 4.92 (1.70)
Valued Living Questionnaire (VLQ) [Mean (Standard Deviation); unit: Composite score on a scale] — The Valued Living Questionnaire (VLQ; Wilson et al., 2010) value and engagement in 10 domains of living. Respondents rate how important each domain is from 1 ("not at all important") to 10 ("extremely important"; Importance subscale) and their engagement in each domain, on a scale from 1 ("not at all consistent with my value") to 10 ("completely consistent with my value"; Consistency subscale). Importance and Consistency scores are multiplied for each domain, added across domains, and then divided by 10 such that possible scores range from 10-100. Higher scores indicate greater valued living. Population: Some participants did not complete or had missing values in this baseline assessment, so the number analyzed is lower than that of the total group.
  Composite score on a scale
    number analyzed (Participants) | 79 | 81 | 160
    (all) | 37.39 (19.42) | 40.72 (16.89) | 39.08 (18.20)

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Impairment Assessed Through the Sheehan Disability Scale (SDS)
Description: The Sheehan Disability Scale (SDS; Sheehan, 1983; Sheehan et al., 1996) is a composite of three self-rated items regarding the degree to which symptoms disrupted work/school, social life, and family life/responsibilities on an 11-point scale ranging from "Not at all" to "Extremely," with an option for "Not applicable". The possible range of scores is 0 to 30. Higher scores indicate greater disability.
Time Frame: Assessments occurred at baseline, every treatment session, post treatment, and approximately 3 and 6 months after post treatment.
Population: The number of participants analyzed differs at the timepoints due to some participants either: 1) not filling out the measure at a given time point due to clinician error; 2) not being present for one of the timepoints; or 3) leaving the study before a given timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Present Centered Therapy: Participants randomized to the PCT arm received 12 sessions of therapy focused on improving day-to-day functioning (with no focus on trauma or re-visiting past experiences). Participants randomized to the PCT arm received 12 sessions of therapy focused on improving day-to-day functioning (with no focus on trauma or re-visiting past experiences). PCT is a manualized evidenced-based PTSD treatment used in several large-scale PTSD trials that focuses on improving functioning. It incorporates the essential therapeutic elements common to different types of psychotherapies, including supportive empathic listening and unconditional positive regard. The therapist plays an active role but does not impart any systematic training. The focus is to create an understanding of how the symptoms of PTSD are related to day-to-day difficulties and to help patients develop new, more adaptive functional responses to these stressors with a problem-focused and problem- solving approach. In prior trials, PCT showed equivalent change to active therapies at the last follow-up. The VA offers PCT as an evidence-based therapy for PTSD.
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 82 | 84
  Baseline | 20.52 (5.14) | 20.43 (5.10)
  Session 1: number analyzed (Participants) | 74 | 77
  Session 1 | 17.39 (5.67) | 18.04 (5.49)
  Session 2: number analyzed (Participants) | 73 | 77
  Session 2 | 16.93 (6.12) | 18.25 (6.47)
  Session 3: number analyzed (Participants) | 70 | 69
  Session 3 | 16.16 (6.45) | 17.36 (6.46)
  Session 4: number analyzed (Participants) | 68 | 70
  Session 4 | 16.16 (7.00) | 17.50 (6.00)
  Session 5: number analyzed (Participants) | 65 | 66
  Session 5 | 14.58 (6.73) | 16.02 (6.97)
  Session 6: number analyzed (Participants) | 65 | 62
  Session 6 | 14.86 (7.27) | 16.16 (7.39)
  Session 7: number analyzed (Participants) | 63 | 62
  Session 7 | 14.33 (6.76) | 15.32 (7.42)
  Session 8: number analyzed (Participants) | 63 | 61
  Session 8 | 12.57 (6.83) | 15.21 (7.03)
  Session 9: number analyzed (Participants) | 58 | 57
  Session 9 | 11.90 (6.54) | 14.16 (7.85)
  Session 10: number analyzed (Participants) | 53 | 52
  Session 10 | 11.51 (6.41) | 13.65 (7.66)
  Session 11: number analyzed (Participants) | 51 | 50
  Session 11 | 11.02 (6.34) | 13.88 (7.42)
  Session 12: number analyzed (Participants) | 51 | 56
  Session 12 | 9.76 (6.44) | 14.04 (7.91)
  3 month follow-up: number analyzed (Participants) | 43 | 52
  3 month follow-up | 13.21 (7.83) | 15.38 (7.71)
  6 month follow-up: number analyzed (Participants) | 37 | 38
  6 month follow-up | 11.22 (6.87) | 15.66 (7.39)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SDS scores, t(1519 )= -2.19, d = 0.15; Test type: Superiority; p = 0.03, Mixed Models Analysis; Slope = -0.236, 95% CI 2-sided [-3.34 to -0.18]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to- treat data for SDS scores, t(160)= -15.74, d = 2.97; Test type: Superiority; p < .001, Mixed Models Analysis; Slope = -8.97, 95% CI 2-sided [-10.12 to -6.11]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SDS scores, t(160) = -12.72, d = 1.86; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -6.62, 95% CI 2-sided [-8.35 to -6.11]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SDS scores, t(1510) = -0.90, d = 0.05; Test type: Superiority; p = 0.49, Mixed Models Analysis; Slope = -0.65, 95% CI 2-sided [-2.13 to 0.86]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for SDS scores, t(1510) = 2.11, d = 0.11; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = 1.10, 95% CI 2-sided [0.06 to 2.17]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SDS scores, t(1510) = 3.45, d = 0.18; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = 1.75, 95% CI 2-sided [0.75 to 2.81]

2. Primary Outcome: Pre-to-Post-Treatment Clinically Significant Change (CSC) in Functional Impairment Assessed Through the Sheehan Disability Scale (SDS)
Description: The investigators used the Jacobson and Truax methodology to index individual participant clinically significant change in functional impairment, assessed through the Sheehan Disability Scale (SDS). Individuals were classified as experiencing probable recovery if they passed the Criterion Cutoff and the RCI criteria; improved if they passed the RCI criterion, but their post-treatment or follow-up score did not pass the Criterion Cutoff; unchanged if they failed to pass the RCI; or deteriorated if they passed the RCI criterion but symptom scores increased.
Time Frame: Baseline and post-treatment.
Population: The participants analyzed here are participants who had a complete SDS baseline assessment, and a complete SDS post-treatment assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 51 | 56
Percentage of participants
  Probable Recovery | 56.86 | 35.71
  Improved | 0 | 12.50
  Unchanged | 43.14 | 48.21
  Deteriorated | 0 | 3.57
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportions of participants who experienced probable recovery in SDS from baseline to post-treatment in AD-MIL versus PCT; Test type: Superiority; p = 0.03, Fisher Exact; Odds Ratio (OR) = 2.35, 95% CI 2-sided [1.01 to 5.56]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportion of participants who experienced improvement from baseline to post-treatment in SDS in AD-MIL versus PCT; Test type: Superiority; p = 0.01, Fisher Exact; Odds Ratio (OR) = 0, 95% CI 2-sided [0 to 0.71]
Statistical Analysis 3: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportion of participants who experienced no change in SDS from baseline to post-treatment in AD-MIL versus PCT; Test type: Superiority; p = .69, Fisher Exact; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.35 to 1.87]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportion of participants who experienced deterioration in SDS from baseline to post-treatment in AD-MIL versus PCT; Test type: Superiority; p = 0.50, Fisher Exact; Odds Ratio (OR) = 0, 0% CI 2-sided [0 to 5.83]

3. Primary Outcome: Change in Psychosocial Functioning Assessed Through the Brief Inventory of Psychosocial Functioning (B-IPF)
Description: The Brief Inventory of Psychosocial Functioning (B-IPF; Marx, 2013) was used to assess functional gains. It is a 7-item scale indexing overall level of functioning in seven life domains: romantic relationship, relationship with children, family relationships, friendships and socializing, work, training and education, and activities of daily living. The investigators used a prorated total percentage for the dimensional ratings, such that Veterans who were not in romantic relationships, had no children, or were not in employed or in school did not have those domains included in their percentage. Possible scores on the B-IPF range from 0% to 100%, with higher scores indicating more issues in psychosocial functioning.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Units on a scale
  Baseline: number analyzed (Participants) | 85 | 82
  Baseline | 59.37 (22.14) | 61.06 (19.38)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 52.68 (25.96) | 55.97 (24.77)
  3 month follow-up: number analyzed (Participants) | 47 | 51
  3 month follow-up | 43.47 (26.98) | 52.87 (28.44)
  6 month follow-up: number analyzed (Participants) | 40 | 39
  6 month follow-up | 41.12 (25.95) | 51.73 (25.31)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for B-IPF scores, t(326) = -0.93, d = 0.10; Test type: Superiority; p = 0.35, Mixed Models Analysis; Slope = -3.39, 95% CI 2-sided [-10.57 to 3.79]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for BIPF scores, t(116) = -3.27, d = 0.61; Test type: Superiority; p = 0.001, Mixed Models Analysis; Slope = -8.64, 95% CI 2-sided [-13.83 to -3.44]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for B-IPF scores, t(116) = -2.08, d = 0.39; Test type: Superiority; p = 0.04, Mixed Models Analysis; Slope = -5.25, 95% CI 2-sided [-10.21 to -0.29]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for B-IPF scores, t(326) = -1.79, d = 0.20; Test type: Superiority; p = 0.08, Mixed Models Analysis; Slope = -5.17, 95% CI 2-sided [-10.86 to 0.52]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for B-IPF scores, t(326) = -2.72, d = 0.30; Test type: Superiority; p = 0.007, Mixed Models Analysis; Slope = -5.64, 95% CI 2-sided [-9.72 to -1.57]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for B-IPF scores, t(326) = -0.23, d = 0.03; Test type: Superiority; p = 0.82, Mixed Models Analysis; Slope = -0.47, 95% CI 2-sided [-4.44 to 3.50]

4. Primary Outcome: Change in Functional Impairment Assessed Through the Sheehan Disability Scale (SDS) for the COVID-19 Cohort
Description: The Sheehan Disability Scale (SDS; Sheehan, 1983; Sheehan et al., 1996) is a composite of three self-rated items regarding the degree to which symptoms disrupted work/school, social life, and family life/responsibilities on an 11-point scale ranging from "Not at all" to "Extremely," with an option for "Not applicable". The investigators used a prorated total mean score for the dimensional ratings such that only social and family ratings will be included for Veterans who were not employed or attending school at the time. The possible range of scores is 0 to 30. Higher scores indicate greater disability.
Time Frame: Assessments occurred at baseline, every treatment session, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 21 | 22
Score on a scale
  Baseline: number analyzed (Participants) | 18 | 22
  Baseline | 21.78 (4.52) | 19.82 (5.83)
  Session 1: number analyzed (Participants) | 18 | 20
  Session 1 | 17.22 (5.07) | 18.15 (4.66)
  Session 2: number analyzed (Participants) | 19 | 20
  Session 2 | 18.47 (5.75) | 19.50 (4.63)
  Session 3: number analyzed (Participants) | 16 | 18
  Session 3 | 16.75 (5.51) | 17.00 (6.56)
  Session 4: number analyzed (Participants) | 17 | 19
  Session 4 | 16.59 (6.56) | 18.00 (5.58)
  Session 5: number analyzed (Participants) | 16 | 18
  Session 5 | 13.00 (5.90) | 14.39 (6.32)
  Session 6: number analyzed (Participants) | 16 | 17
  Session 6 | 12.88 (4.98) | 16.24 (5.27)
  Session 7: number analyzed (Participants) | 15 | 18
  Session 7 | 13.53 (5.85) | 14.22 (6.32)
  Session 8: number analyzed (Participants) | 15 | 17
  Session 8 | 13.73 (5.26) | 14.06 (5.40)
  Session 9: number analyzed (Participants) | 14 | 18
  Session 9 | 11.29 (5.11) | 12.67 (6.64)
  Session 10: number analyzed (Participants) | 13 | 17
  Session 10 | 10.77 (4.51) | 13.00 (8.06)
  Session 11: number analyzed (Participants) | 14 | 17
  Session 11 | 9.93 (5.28) | 11.53 (7.21)
  Session 12: number analyzed (Participants) | 13 | 17
  Session 12 | 9.08 (5.94) | 13.18 (7.99)
  3 month follow-up: number analyzed (Participants) | 3 | 9
  3 month follow-up | 19.00 (5.29) | 15.56 (7.06)
  6 month follow-up: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SDS scores for the COVID-19 cohort, t(373) = -0.32, d = 0.03; Test type: Superiority; p = 0.75, Mixed Models Analysis; Slope = -0.60, 95% CI 2-sided [-4.68 to 3.36]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for SDS scores for the COVID-19 cohort, t(37) = -6.01, d = 1.97; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -9.12, 95% CI 2-sided [-12.12 to -6.12]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SDS scores for the COVID-19 cohort, t(37) = -6.11, d = 2.01; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -8.72, 95% CI 2-sided [-11.16 to -5.76]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SDS scores for the COVID-19 cohort, t(373) = -0.59, d = 0.06; Test type: Superiority; p = 0.56, Mixed Models Analysis; Slope = -2.28, 95% CI 2-sided [-10.08 to 5.52]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for SDS scores for the COVID-19 cohort, t(373) = 1.25, d = 0.13; Test type: Superiority; p = 0.22, Mixed Models Analysis; Slope = 4.20, 95% CI 2-sided [-0.24 to 10.92]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SDS scores for the COVID-19 cohort, t(373) = 3.18, d = 0.33; Test type: Superiority; p = 0.002, Mixed Models Analysis; Slope = 6.60, 95% CI 2-sided [2.52 to 10.69]

5. Primary Outcome: Change in PTSD Symptom Burden Assessed Through the PTSD Checklist for DSM-5 (PCL-5) for the COVID-19 Cohort
Description: The PTSD Checklist for DSM-5 (PCL-5; Weathers et al., 2013) is a 20-item self-report checklist based on the 20 DSM-5 symptoms post-traumatic stress disorder (PTSD). The PCL-5 has been validated as a means of monitoring symptom change during treatment. The 20 items are scored are scored in the past month on a scale from 0 ("not at all") to 4 ("extremely"), generating a total symptom severity score between 0 and 80, with higher scores indicating greater PTSD symptom severity.
Time Frame: Assessments occurred at baseline, every treatment session, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 21 | 22
Score on a scale
  Baseline: number analyzed (Participants) | 15 | 20
  Baseline | 48.53 (8.84) | 50.62 (11.57)
  Session 1: number analyzed (Participants) | 18 | 20
  Session 1 | 47.11 (12.07) | 46.48 (10.87)
  Session 2: number analyzed (Participants) | 19 | 20
  Session 2 | 41.65 (11.33) | 47.15 (12.73)
  Session 3: number analyzed (Participants) | 17 | 18
  Session 3 | 43.24 (13.10) | 45.22 (10.11)
  Session 4: number analyzed (Participants) | 17 | 19
  Session 4 | 42.47 (13.68) | 45.89 (8.81)
  Session 5: number analyzed (Participants) | 16 | 18
  Session 5 | 40.50 (17.04) | 39.72 (12.21)
  Session 6: number analyzed (Participants) | 16 | 17
  Session 6 | 36.75 (15.26) | 42.00 (10.81)
  Session 7: number analyzed (Participants) | 15 | 18
  Session 7 | 36.40 (12.20) | 37.78 (12.83)
  Session 8: number analyzed (Participants) | 15 | 17
  Session 8 | 33.67 (12.11) | 37.47 (14.69)
  Session 9: number analyzed (Participants) | 14 | 18
  Session 9 | 30.50 (13.14) | 37.44 (13.43)
  Session 10: number analyzed (Participants) | 13 | 17
  Session 10 | 31.69 (14.29) | 35.53 (14.89)
  Session 11: number analyzed (Participants) | 14 | 17
  Session 11 | 30.14 (14.72) | 35.29 (14.55)
  Session 12: number analyzed (Participants) | 13 | 17
  Session 12 | 29.15 (12.11) | 37.47 (14.49)
  3-month follow-up: number analyzed (Participants) | 3 | 9
  3-month follow-up | 30.33 (11.59) | 40.47 (20.46)
  6-month follow-up: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PCL-5 scores for the COVID-19 cohort, t(367) = 0.10, d = 0.01; Test type: Superiority; p = 0.92, Mixed Models Analysis; Slope = 0.48, 95% CI 2-sided [-9.60 to 10.69]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for PCL-5 scores for the COVID-19 cohort, t(37) = -4.23, d = 1.39; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -16.08, 95% CI 2-sided [-23.64 to -8.52]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PCL-5 scores for the COVID-19 cohort, t(37) = -4.77, d = 1.57; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -16.56, 95% CI 2-sided [-23.40 to -9.72]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PCL-5 scores for the COVID-19 cohort, t(367) = -3.15, d = 0.33; Test type: Superiority; p = 0.002, Mixed Models Analysis; Slope = -26.28, 95% CI 2-sided [-42.60 to -9.84]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for PCL-5 scores for the COVID-19 cohort, t(37) = -2.67, d = 0.28; Test type: Superiority; p = 0.01, Mixed Models Analysis; Slope = -18.72, 95% CI 2-sided [-32.40 to -4.92]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for B- IPF scores, the Pre-Post PCT Time slope was -5.25 [95% CI = -10.21, -0.29], p-value = 0.04, t(116) = -2.08, d = 0.39; Test type: Superiority; p = 0.04, Mixed Models Analysis; Slope = -5.25, 95% CI 2-sided [-10.21 to -0.29]

6. Primary Outcome: Change in PTSD Symptom Severity and Diagnosis Assessed Through the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) for the COVID-19 Cohort
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5; Weathers et al., 2013) is closely modeled on the CAPS-IV, a structured diagnostic interview and gold standard for assessing PTSD. It has excellent psychometric properties and diagnostic efficiency (Weathers et al., 2001). The CAPS-5 uses a single 4-point ordinal rating scale to measure symptom severity. These ratings combine information about symptom frequency and intensity obtained by the interviewer. CAPS-5 scores range from 0 to 80, with higher scores indicating greater PTSD symptom severity.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 21 | 22
Score on a scale
  Baseline | 39.76 (8.89) | 40.86 (9.15)
  Post treatment: number analyzed (Participants) | 14 | 19
  Post treatment | 24.07 (13.51) | 34.79 (11.92)
  3 month follow-up: number analyzed (Participants) | 6 | 9
  3 month follow-up | 35.50 (7.82) | 28.33 (17.63)
  6 month follow-up: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CAPS-5 scores for the COVID-19 cohort, t(49) = -1.69, d = 0.48; Test type: Superiority; p = 0.10, Mixed Models Analysis; Slope = -6.38, 95% CI 2-sided [-13.97 to 1.22]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for CAPS-5 scores for the COVID-19 cohort, t(32) = -4.71, d = 1.67; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -13.29, 95% CI 2-sided [-18.96 to -7.62]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CAPS-5 scores for the COVID-19 cohort, t(32) = -2.75, d = 0.97; Test type: Superiority; p = 0.001, Mixed Models Analysis; Slope = -6.92, 95% CI 2-sided [-11.96 to -1.87]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CAPS-5 scores for the COVID-19 cohort, t(49) = 0.97, d = 0.28; Test type: Superiority; p = 0.34, Mixed Models Analysis; Slope = 5.22, 95% CI 2-sided [-5.60 to 16.05]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for CAPS-5 scores for the COVID-19 cohort, t(49) = 1.40, d = 0.40; Test type: Superiority; p = 0.17, Mixed Models Analysis; Slope = 5.93, 95% CI 2-sided [-2.55 to 14.41]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CAPS-5 scores for the COVID-19 cohort, t(49) = 0.21, d = 0.06; Test type: Superiority; p = 0.83, Mixed Models Analysis; Slope = 0.70, 95% CI 2-sided [-6.04 to 7.44]

7. Primary Outcome: Change in Symptoms of Depression Assessed Through the Patient Health Questionnaire (PHQ-9) for the COVID-19 Cohort
Description: The Patient Health Questionnaire (PHQ-9) is widely used and well-validated measure of symptoms of depression (Kroenke et al., 2001). It scores each of the nine DSM criteria for depression on a scale of 0 ("not at all") to 3 ("nearly every day"). The range of possible scores is 0 to 27. A higher score indicates more frequent depression symptoms.
Time Frame: Assessments occurred at baseline, every treatment session, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 21 | 22
Score on a scale
  Baseline: number analyzed (Participants) | 13 | 20
  Baseline | 17.31 (5.38) | 14.95 (6.14)
  Session 1: number analyzed (Participants) | 18 | 20
  Session 1 | 15.07 (6.37) | 16.14 (4.13)
  Session 2: number analyzed (Participants) | 18 | 20
  Session 2 | 14.44 (5.87) | 16.02 (5.08)
  Session 3: number analyzed (Participants) | 17 | 18
  Session 3 | 13.79 (4.95) | 15.56 (5.43)
  Session 4: number analyzed (Participants) | 17 | 19
  Session 4 | 13.82 (5.44) | 14.92 (4.08)
  Session 5: number analyzed (Participants) | 16 | 18
  Session 5 | 15.10 (5.05) | 12.28 (4.12)
  Session 6: number analyzed (Participants) | 16 | 17
  Session 6 | 12.60 (6.08) | 12.37 (3.47)
  Session 7: number analyzed (Participants) | 15 | 18
  Session 7 | 12.40 (6.73) | 11.90 (4.56)
  Session 8: number analyzed (Participants) | 15 | 17
  Session 8 | 12.27 (6.38) | 12.46 (4.93)
  Session 9: number analyzed (Participants) | 14 | 18
  Session 9 | 11.20 (5.45) | 12.78 (5.92)
  Session 10: number analyzed (Participants) | 13 | 17
  Session 10 | 11.86 (7.15) | 12.59 (5.42)
  Session 11: number analyzed (Participants) | 14 | 17
  Session 11 | 10.56 (5.77) | 11.84 (4.69)
  Session 12: number analyzed (Participants) | 13 | 17
  Session 12 | 10.47 (5.21) | 11.53 (4.61)
  3 month follow-up: number analyzed (Participants) | 3 | 9
  3 month follow-up | 18.00 (7.55) | 14.10 (6.02)
  6 month follow-up: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PHQ-9 scores for the COVID-19 cohort, t(373) = 0.30, d = 0.03; Test type: Superiority; p = 0.76, Mixed Models Analysis; Slope = 0.60, 95% CI 2-sided [-3.12 to 4.20]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for PHQ-9 scores for the COVID-19 cohort, t(37) = -3.14, d = 1.03; Test type: Superiority; p = 0.002, Mixed Models Analysis; Slope = -3.12, 95% CI 2-sided [-6.96 to -1.56]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PHQ-9 scores for the COVID-19 cohort, t(37) = -3.88, d = 1.27; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -4.92, 95% CI 2-sided [-7.32 to -2.40]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PHQ-9 scores for the COVID-19 cohort, t(373) = -1.50, d = 0.16; Test type: Superiority; p = 0.13, Mixed Models Analysis; Slope = -4.80, 95% CI 2-sided [-11.16 to 1.44]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for PHQ-9 scores for the COVID-19 cohort, t(373) = -0.87, d = 0.09; Test type: Superiority; p = 0.38, Mixed Models Analysis; Slope = -2.40, 95% CI 2-sided [-7.68 to 3.00]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PHQ-9 scores for the COVID-19 cohort, t(373) = 1.42, d = 0.15; Test type: Superiority; p = 0.26, Mixed Models Analysis; Slope = 2.40, 95% CI 2-sided [-0.96 to 5.88]

8. Secondary Outcome: Change in PTSD Symptom Severity and Diagnosis Assessed Through the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
Description: as for outcome 6
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Adaptive Disclosure for Moral Injury and Loss: AD-MIL is a 12-session treatment designed to address shame and guilt and to develop compassion for the self and the other. At the outset of AD-MIL, the investigators ask Veterans to enlist a family member or friend to provide support and to reinforce their plan for adaptive, purposeful functioning moving forward. The sessions that follow homework assignments involve a discussion to reinforce positive steps taken and identifying obstacles to completion (e.g., self-defeating beliefs). There is a special emphasis on discussing self-handicapping, namely feeling unworthy of getting better or living a good life. The goal is not only for Veterans to develop a sense of mastery in accomplishing tasks and to experience the benefits of the activities, but also to work on overcoming feelings of unworthiness.
- Present Centered Therapy: PCT is a manualized evidenced-based PTSD treatment used in several large-scale PTSD trials. It incorporates the essential therapeutic elements common to different types of psychotherapies, including supportive empathic listening and unconditional positive regard. The therapist plays an active role, but does not impart any systematic training. The focus is to create an understanding of how the symptoms of PTSD are related to day-to-day difficulties and to help patients develop new, more adaptive responses to these stressors with a problem-focused and problem-solving approach. In prior trials, PCT showed equivalent change to active therapies at the last follow-up. The VA offers PCT as an evidence-based therapy for PTSD.
  Present Centered Therapy: Participants randomized to the PCT arm will receive 12 sessions of therapy focused on problems occurring in the present (with no focus on trauma or re-visiting past experiences).
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline | 36.08 (11.88) | 35.69 (13.60)
  Post treatment: number analyzed (Participants) | 59 | 66
  Post treatment | 21.78 (14.92) | 30.74 (12.41)
  3 month follow-up: number analyzed (Participants) | 54 | 52
  3 month follow-up | 24.44 (14.37) | 29.63 (13.68)
  6 month follow-up: number analyzed (Participants) | 43 | 41
  6 month follow-up | 21.16 (15.47) | 27.41 (13.07)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CAPS-5 scores, t(348) = -3.65, d = 0.39; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -6.65, 95% CI 2-sided [-10.23 to -3.07]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for CAPS-5 scores, t(131) = -9.14, d = 1.60; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -11.88, 95% CI 2-sided [-14.43 to -9.32]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CAPS-5 scores, t(131) = -4.10, d = 0.72; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -5.23, 95% CI 2-sided [-7.74 to -2.72]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CAPS-5 scores, t(348) = 0.87, d = 0.09; Test type: Superiority; p = 0.39, Mixed Models Analysis; Slope = 1.36, 95% CI 2-sided [-1.73 to 4.45]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for CAPS-5 scores, t(348) = 0.07, d = 0.001; Test type: Superiority; p = 0.94, Mixed Models Analysis; Slope = 0.08, 95% CI 2-sided [-2.10 to 2.26]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CAPS-5 scores, t(348) = -1.15, d = 0.12; Test type: Superiority; p = 0.25, Mixed Models Analysis; Slope = -1.28, 95% CI 2-sided [-3.48 to 0.91]

9. Secondary Outcome: Pre- to Post-Treatment Clinically Significant Change (CSC) in PTSD Symptom Severity and Diagnosis Assessed Through the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
Description: The investigators used the Jacobson and Truax methodology to index individual participant clinically significant change in PTSD symptom severity and diagnosis, which the investigators assessed through the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). Individuals were classified as experiencing probable recovery if they passed the Criterion Cutoff and the RCI criteria; improved if they passed the RCI criterion, but their post-treatment or follow-up score did not pass the Criterion Cutoff; unchanged if they failed to pass the RCI; or deteriorated if they passed the RCI criterion but symptom scores increased.
Time Frame: Baseline and post treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 59 | 66
Percentage of participants
  Probable Recovery | 15.25 | 3.03
  Improved | 30.51 | 25.76
  Unchanged | 52.54 | 63.64
  Deteriorated | 1.69 | 10.61
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportions of participants who experienced probable recovery in CAPS-5 from baseline to post-treatment in AD-MIL versus PCT; Test type: Superiority; p = 0.01, Fisher Exact; Odds Ratio (OR) = 6.44, 95% CI 2-sided [1.29 to 63.18]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportions of participants who experienced improvement in CAPS-5 from baseline to post-treatment in AD-MIL versus PCT; Test type: Superiority; p = 0.40, Fisher Exact; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.61 to 3.75]
Statistical Analysis 3: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportions of participants who experienced no change in CAPS-5 from baseline to post-treatment in AD-MIL versus PCT; Test type: Superiority; p = 0.58, Fisher Exact; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.36 to 1.70]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportions of participants who experienced deterioration in CAPS-5 from baseline to post-treatment in AD-MIL versus PCT; Test type: Superiority; p = 0.06, Fisher Exact; Odds Ratio (OR) = 0.15, 95% CI 2-sided [0.003 to 1.20]

10. Secondary Outcome: Change in PTSD Caseness Assessed Through PTSD Diagnoses Using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5; Weathers et al., 2013) is closely modeled on the CAPS-IV, a structured diagnostic interview and gold standard for assessing PTSD. It has excellent psychometric properties and diagnostic efficiency (Weathers et al., 2001). The CAPS-5 uses a single 4-point ordinal rating scale to measure symptom severity. These ratings combine information about symptom frequency and intensity obtained by the interviewer. A patient is determined to have met the DSM-5 criteria for PTSD if they have endorsed at least one symptom from the B cluster, at least one symptom from the C Cluster, and at least two symptoms from the E cluster, along with experiencing the symptoms for at least one month and reporting clinically significant distress or functional impairment.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: The number of participants analyzed differs at the timepoints due to some participants either 1) not filling out the measure at a given time point due to clinician error or 2) leaving the study before a given timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- Adaptive Disclosure for Moral Injury and Loss: AD-MIL is a manualized 12-session individual psychotherapy designed to improve functioning and to reduce PTSD symptoms by facilitating Veterans doing corrective things in their life to heal and repair traumatic loss and moral injuries. The change agents are: (1) emotional-processing of traumatic loss and moral injuries and motivating a healing and action plan by writing therapeutic letters (e.g., to a lost unit member, to victims of personal transgressions, to people who transgressed); (2) skills training and behavioral contracting to improve functioning and targeting moral injury- and traumatic loss-related psychological and behavioral obstacles to positive and potentially habilitative engagements in occupational, relationship, and family roles; and (3) teaching self- and other-compassion and mindfulness. The goal is to redress the functional impact of moral emotions (anger, shame).
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Participants
  Baseline | 89 | 85
  Post treatment: number analyzed (Participants) | 59 | 66
  Post treatment | 30 | 45
  3 month follow-up: number analyzed (Participants) | 54 | 52
  3 month follow-up | 31 | 35
  6 month follow-up: number analyzed (Participants) | 42 | 41
  6 month follow-up | 19 | 27
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportions of participants with a PTSD Diagnosis in CAPS-5 at post-treatment in AD-MIL versus PCT; Test type: Superiority; p = 0.07, Fisher Exact; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.22 to 1.06]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportions of participants with PTSD Diagnosis in CAPS-5 at 3MFU in AD-MIL versus PCT; Test type: Superiority; p = 0.33, Fisher Exact; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.28 to 1.56]
Statistical Analysis 3: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportions of participants with PTSD Diagnosis in CAPS-5 at 6MFU in AD-MIL versus PCT; Test type: Superiority; p = 0.05, Fisher Exact; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.15 to 1.08]

11. Secondary Outcome: Change in PTSD Symptom Burden Assessed Through the PTSD Checklist for DSM-5 (PCL-5)
Description: as for outcome 5
Time Frame: Assessments occurred at baseline, every treatment session, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 83 | 83
  Baseline | 49.26 (11.43) | 51.66 (10.85)
  Session 1: number analyzed (Participants) | 76 | 78
  Session 1 | 45.79 (13.24) | 45.60 (12.72)
  Session 2: number analyzed (Participants) | 74 | 76
  Session 2 | 42.49 (13.91) | 44.01 (13.60)
  Session 3: number analyzed (Participants) | 72 | 70
  Session 3 | 42.46 (13.88) | 42.81 (13.76)
  Session 4: number analyzed (Participants) | 70 | 71
  Session 4 | 42.06 (14.36) | 42.68 (12.83)
  Session 5: number analyzed (Participants) | 67 | 67
  Session 5 | 41.08 (16.14) | 40.23 (14.53)
  Session 6: number analyzed (Participants) | 66 | 63
  Session 6 | 38.42 (15.40) | 38.72 (14.34)
  Session 7: number analyzed (Participants) | 64 | 63
  Session 7 | 36.64 (15.21) | 38.43 (14.06)
  Session 8: number analyzed (Participants) | 64 | 61
  Session 8 | 33.48 (15.67) | 37.76 (15.83)
  Session 9: number analyzed (Participants) | 59 | 58
  Session 9 | 31.83 (16.63) | 35.40 (15.53)
  Session 10: number analyzed (Participants) | 53 | 53
  Session 10 | 30.51 (16.80) | 34.32 (15.25)
  Session 11: number analyzed (Participants) | 52 | 50
  Session 11 | 29.37 (16.44) | 34.82 (15.51)
  Session 12: number analyzed (Participants) | 56 | 55
  Session 12 | 27.33 (15.78) | 35.48 (15.72)
  3 month follow-up: number analyzed (Participants) | 46 | 52
  3 month follow-up | 29.88 (18.61) | 38.40 (15.63)
  6 month follow-up: number analyzed (Participants) | 39 | 39
  6 month follow-up | 31.43 (18.80) | 35.79 (15.90)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PCL-5 scores, t(1542) = -3.01, d = 0.13; Test type: Superiority; p = .003, Mixed Models Analysis; Slope = -4.63, 95% CI 2-sided [-7.16 to -2.10]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for PCL-5 scores, t(161) = -11.50, d = 1.81; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -12.62, 95% CI 2-sided [-14.43 to -10.80]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PCL-5 scores, t(161) = -7.40, d = 1.16; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -7.89, 95% CI 2-sided [-9.77 to -6.20]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PCL-5 scores, t(1542) = -0.45, d = 0.02; Test type: Superiority; p = 0.65, Mixed Models Analysis; Slope = -0.75, 95% CI 2-sided [-4.01 to 2.52]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for PCL-5 scores, t(1542) = 1.94, d = 0.10; Test type: Superiority; p = 0.05, Mixed Models Analysis; Slope = 2.30, 95% CI 2-sided [-0.03 to 4.63]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PCL-5 scores, t(1542) = 2.61, d = 0.13; Test type: Superiority; p = 0.001, Mixed Models Analysis; Slope = 3.04, 95% CI 2-sided [0.75 to 5.34]

12. Secondary Outcome: Pre- to Post-Treatment Clinically Significant Change (CSC) in PTSD Symptom Burden Assessed Through the PTSD Checklist for DSM-5 (PCL-5)
Description: The investigators used the Jacobson and Truax methodology to index individual participant clinically significant change in PTSD symptom burden, which the investigators assessed through the PTSD Checklist for DSM-5 (PCL-5). Individuals were classified as experiencing probable recovery if they passed the Criterion Cutoff and the RCI criteria; improved if they passed the RCI criterion, but their post-treatment or follow-up score did not pass the Criterion Cutoff; unchanged if they failed to pass the RCI; or deteriorated if they passed the RCI criterion but symptom scores increased.
Time Frame: Baseline and post treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 56 | 55
Percentage of participants
  Probable Recovery | 42.86 | 25.45
  Improved | 17.86 | 23.64
  Unchanged | 37.50 | 50.91
  Deteriorated | 1.79 | 0
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportions of participants experiencing probable recovery in PCL-5 at post-treatment in AD-MIL versus PCT; Test type: Superiority; p = 0.04, Fisher Exact; Odds Ratio (OR) = 2.39, 95% CI 2-sided [1.01 to 5.84]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportions of participants experiencing improvement in PCL-5 at post-treatment in AD-MIL versus PCT; Test type: Superiority; p = 0.49, Fisher Exact; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.25 to 1.95]
Statistical Analysis 3: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; Odds ratio comparison of the proportions of participants experiencing no change in PCL-5 at post-treatment in AD-MIL versus PCT; Test type: Superiority; p = 0.18, Fisher Exact; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.25 to 1.32]

13. Secondary Outcome: Change in Symptoms of Depression Assessed Through the Patient Health Questionnaire (PHQ-9)
Description: as for outcome 7
Time Frame: Assessments occurred at baseline, every treatment session, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 79 | 82
  Baseline | 16.88 (5.43) | 16.62 (5.50)
  Session 1: number analyzed (Participants) | 76 | 79
  Session 1 | 15.92 (6.05) | 15.70 (5.44)
  Session 2: number analyzed (Participants) | 73 | 78
  Session 2 | 14.80 (5.60) | 15.81 (5.55)
  Session 3: number analyzed (Participants) | 72 | 70
  Session 3 | 14.56 (5.43) | 15.14 (5.83)
  Session 4: number analyzed (Participants) | 70 | 70
  Session 4 | 14.47 (5.54) | 14.95 (5.03)
  Session 5: number analyzed (Participants) | 67 | 67
  Session 5 | 14.53 (5.74) | 14.30 (5.87)
  Session 6: number analyzed (Participants) | 66 | 63
  Session 6 | 13.85 (6.43) | 13.26 (5.25)
  Session 7: number analyzed (Participants) | 64 | 63
  Session 7 | 12.89 (6.20) | 13.19 (5.73)
  Session 8: number analyzed (Participants) | 64 | 61
  Session 8 | 12.34 (6.91) | 13.32 (5.99)
  Session 9: number analyzed (Participants) | 59 | 58
  Session 9 | 11.47 (6.18) | 12.67 (6.11)
  Session 10: number analyzed (Participants) | 54 | 53
  Session 10 | 11.26 (6.92) | 12.05 (5.90)
  Session 11: number analyzed (Participants) | 52 | 51
  Session 11 | 11.17 (6.22) | 12.29 (6.07)
  Session 12: number analyzed (Participants) | 56 | 56
  Session 12 | 9.99 (6.30) | 11.56 (5.75)
  3 month follow-up: number analyzed (Participants) | 46 | 51
  3 month follow-up | 12.22 (7.61) | 14.17 (6.29)
  6 month follow-up: number analyzed (Participants) | 38 | 39
  6 month follow-up | 11.84 (7.14) | 13.15 (7.28)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PHQ-9 scores, t(1550) = -1.46, d = 0.07; Test type: Superiority; p = 0.14, Mixed Models Analysis; Slope = -0.99, 95% CI 2-sided [-2.29 to 0.34]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for PHQ-9 scores, t(161) = -12.41, d = 1.96; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -5.87, 95% CI 2-sided [-6.80 to -4.90]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PHQ-9 scores, t(161) = -10.29, d = 1.62; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -4.89, 95% CI 2-sided [-5.82 to -3.94]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PHQ-9 scores, t(1550) = 0.42, d = 0.02; Test type: Superiority; p = 0.68, Mixed Models Analysis; Slope = 0.02, 95% CI 2-sided [-0.99 to 1.53]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for PHQ-9 scores, t(1550) = 3.02, d = 0.15; Test type: Superiority; p = 0.003, Mixed Models Analysis; Slope = 1.36, 95% CI 2-sided [0.48 to 2.24]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for PHQ-9 scores, t(1550) = 2.37, d = 0.12; Test type: Superiority; p = 0.02, Mixed Models Analysis; Slope = 1.09, 95% CI 2-sided [0.19 to 1.99]

14. Secondary Outcome: Change in Guilt Cognitions About a Specific Warzone Event Assessed Through the (Lack of) Justification Subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief)
Description: The (lack of) Justification subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief; Kubany et al., 1996) is a 4-item measure that assesses guilty thoughts about the justification of one's actions related to a specific traumatic event. Possible scores range from 0 to 4, with higher scores indicating increased guilt.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 81 | 80
  Baseline | 1.88 (0.98) | 2.00 (0.96)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 1.59 (0.92) | 1.86 (1.10)
  3 month follow-up: number analyzed (Participants) | 46 | 52
  3 month follow-up | 1.70 (1.06) | 2.08 (1.12)
  6 month follow-up: number analyzed (Participants) | 40 | 39
  6 month follow-up | 1.87 (1.26) | 1.78 (1.21)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRGI Justification scores, t(314) = -1.35, d = 0.15; Test type: Superiority; p = 0.18, Mixed Models Analysis; Slope = -0.20, 95% CI 2-sided [-0.49 to 0.09]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for TRGI Justification scores, t(113) = -2.44, d = 0.46; Test type: Superiority; p = 0.02, Mixed Models Analysis; Slope = -0.26, 95% CI 2-sided [-0.47 to -0.05]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRGI Justification scores, t(113) = -0.69, d = 0.12; Test type: Superiority; p = 0.62, Mixed Models Analysis; Slope = -0.06, 95% CI 2-sided [-0.26 to 0.14]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRGI Justification scores, t(314) = 1.34, d = 0.15; Test type: Superiority; p = 0.18, Mixed Models Analysis; Slope = 0.16, 95% CI 2-sided [-0.07 to 0.39]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for TRGI Justification scores, t(113) = 1.49, d = 0.28; Test type: Superiority; p = 0.14, Mixed Models Analysis; Slope = 0.13, 95% CI 2-sided [-0.04 to 0.30]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRGI Justification scores, t(113) = -0.38, d = 0.07; Test type: Superiority; p = 0.71, Mixed Models Analysis; Slope = -0.03, 95% CI 2-sided [-0.19 to 0.13]

15. Secondary Outcome: Change in Guilt Cognitions About a Specific Warzone Event Assessed Through the Hindsight-Bias Subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief)
Description: The Hindsight-Bias subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief; Kubany et al., 1996) is a 7-item measure that assesses guilty thoughts about the preventability and responsibility of a traumatic event. Possible scores range from 0 to 4, with higher scores indicating increased guilt.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 81 | 80
  Baseline | 1.66 (1.06) | 1.68 (1.04)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 0.93 (0.95) | 1.51 (1.05)
  3 month follow-up: number analyzed (Participants) | 46 | 52
  3 month follow-up | 0.98 (1.08) | 1.31 (1.15)
  6 month follow-up: number analyzed (Participants) | 40 | 39
  6 month follow-up | 1.13 (1.24) | 1.09 (0.83)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRGI Hindsight-Bias scores, t(314) = -3.41, d = 0.39; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -0.47, 95% CI 2-sided [-0.74 to -0.20]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for TRGI Hindsight-Bias scores, t(113) = -6.41, d = 1.20; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -0.64, 95% CI 2-sided [-0.83 to -0.44]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRGI Hindsight-Bias scores, t(113) = -1.83, d = 0.34; Test type: Superiority; p = 0.07, Mixed Models Analysis; Slope = -0.17, 95% CI 2-sided [-0.36 to 0.02]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRGI Hindsight-Bias scores, t(314) = 3.13, d = 0.06; Test type: Superiority; p = 0.002, Mixed Models Analysis; Slope = 0.35, 95% CI 2-sided [0.13 to 0.57]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for TRGI Hindsight-Bias scores, t(113) = 2.21, d = 0.42; Test type: Superiority; p = 0.03, Mixed Models Analysis; Slope = 0.18, 95% CI 2-sided [0.02 to 0.34]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRGI Hindsight-Bias scores, t(113) = -2.22, d = 0.42; Test type: Superiority; p = 0.03, Mixed Models Analysis; Slope = -0.17, 95% CI 2-sided [-0.32 to -0.02]

16. Secondary Outcome: Change in Guilt Cognitions About a Specific Warzone Event Assessed Through the Wrongdoing Subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief)
Description: The Wrongdoing subscale of the Brief Trauma Related Guilt Inventory (TRGI-Brief; Kubany et al., 1996) is a 5-item measure that assesses guilty thoughts about wrongdoing tied to a specific traumatic event. Possible scores range from 0 to 4, with higher scores indicating increased guilt.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 81 | 80
  Baseline | 1.71 (1.00) | 1.74 (1.01)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 1.34 (0.95) | 1.65 (1.03)
  3 month follow-up: number analyzed (Participants) | 46 | 52
  3 month follow-up | 1.33 (0.97) | 1.51 (1.04)
  6 month follow-up: number analyzed (Participants) | 40 | 39
  6 month follow-up | 1.42 (1.06) | 1.29 (0.93)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRGI Wrongdoing scores, t(314) = 2.46, d = 0.28; Test type: Superiority; p = 0.01, Mixed Models Analysis; Slope = 0.32, 95% CI 2-sided [0.06 to 0.57]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for RGI Wrongdoing scores, t(113) = 0.06, d = 0.01; Test type: Superiority; p = 0.95, Mixed Models Analysis; Slope = 0.001, 95% CI 2-sided [-0.17 to 0.18]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for RGI Wrongdoing scores, t(113) = -3.32, d = 0.62; Test type: Superiority; p = 0.01, Mixed Models Analysis; Slope = -0.31, 95% CI 2-sided [-0.50 to -0.13]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRGI Wrongdoing scores, t(314) = -2.02, d = 0.23; Test type: Superiority; p = 0.04, Mixed Models Analysis; Slope = -0.21, 95% CI 2-sided [-0.41 to -0.01]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for TRGI Wrongdoing scores, t(113) = -2.18, d = 0.03; Test type: Superiority; p = 0.03, Mixed Models Analysis; Slope = -0.16, 95% CI 2-sided [-0.30 to -0.02]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for RGI Wrongdoing scores, t(113) = 0.70, d = 0.13; Test type: Superiority; p = 0.48, Mixed Models Analysis; Slope = 0.05, 95% CI 2-sided [-0.09 to 0.20]

17. Secondary Outcome: Change in Shame Tied to a Specific Warzone Event Assessed Through the Internal Shame Subscale of the Trauma-Related Shame Inventory (TRSI)
Description: The Internal Shame Subscale of the Trauma-Related Shame Inventory (TRSI; Øktedalen et al., 2014) is a 12-item self-report instrument designed to assess individuals' negative self-evaluations in the context of their traumatic experiences. Possible scores range from 0 to 36, with higher scores indicating more negative self-evaluations. The measure has demonstrated good construct validity (Øktedalen et al., 2014).
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 82 | 80
  Baseline | 12.74 (7.94) | 14.23 (9.46)
  Post treatment: number analyzed (Participants) | 48 | 59
  Post treatment | 11.71 (8.66) | 12.76 (8.31)
  3 month follow-up: number analyzed (Participants) | 46 | 52
  3 month follow-up | 10.59 (8.36) | 12.00 (8.68)
  6 month follow-up: number analyzed (Participants) | 40 | 39
  6 month follow-up | 10.56 (6.69) | 11.69 (6.70)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRSI scores, t(317) = 0.76, d = 0.09; Test type: Superiority; p = 0.45, Mixed Models Analysis; Slope = 0.70, 95% CI 2-sided [-1.12 to 2.52]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for TRSI scores, t(113) = -1.79, d = 0.34; Test type: Superiority; p = 0.08, Mixed Models Analysis; Slope = -1.20, 95% CI 2-sided [-2.52 to 0.12]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRSI scores, t(113) = -3.00, d = 0.56; Test type: Superiority; p = 0.003, Mixed Models Analysis; Slope = -1.91, 95% CI 2-sided [-3.15 to -0.66]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for TRSI scores, t(317) = -0.39, d = 0.04; Test type: Superiority; p = 0.70, Mixed Models Analysis; standardized effect size of the slope = -0.29, 95% CI 2-sided [-1.75 to 1.17]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for TRSI scores, t(317) = -1.11, d = 0.12; Test type: Superiority; p = 0.27, Mixed Models Analysis; Slope = -0.59, 95% CI 2-sided [-1.64 to 0.46]
Statistical Analysis 6: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for TRSI scores, t(317) = -0.57, d = 0.06; Test type: Superiority; p = 0.57, Mixed Models Analysis; Slope = -0.29, 95% CI 2-sided [-1.32 to 0.72]

18. Secondary Outcome: Change in Psychological Health and Distress Assessed Through the Schwartz Outcome Scale-10 (SOS-10)
Description: The Schwartz Outcome Scale-10 (SOS-10; Blais et al., 1999) is a 10-item general mental health outcome measure meant to capture psychological health and distress. Possible scores range from 0 to 60 with higher scores indicating better psychological health and lower distress. The SOS-10 has demonstrated good psychometric properties (Blais et al., 1999).
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 85 | 82
  Baseline | 24.94 (9.87) | 25.43 (8.38)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 32.16 (12.72) | 29.53 (11.18)
  3 month follow-up: number analyzed (Participants) | 47 | 51
  3 month follow-up | 32.43 (13.23) | 26.78 (10.75)
  6 month follow-up: number analyzed (Participants) | 40 | 39
  6 month follow-up | 31.98 (13.37) | 28.85 (11.60)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SOS-10 scores, t(326) = 2.35, d = 0.26; Test type: Superiority; p = 0.02, Mixed Models Analysis; Slope = 3.41, 95% CI 2-sided [0.56 to 6.25]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for SOS-10 scores, t(116) = -6.53, d = 1.21; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = 6.84, 95% CI 2-sided [4.78 to 8.90]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SOS-10 scores, t(116) = 3.44, d = 0.64; Test type: Superiority; p = 0.001, Mixed Models Analysis; Slope = 3.43, 95% CI 2-sided [1.47 to 5.40]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SOS-10 scores, t(326) = 0.66, d = 0.07; Test type: Superiority; p = 0.51, Mixed Models Analysis; Slope = 0.76, 95% CI 2-sided [-1.50 to 3.03]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for SOS-10 scores, t(326) = -0.32, d = 0.04; Test type: Superiority; p = 0.75, Mixed Models Analysis; Slope = -0.27, 95% CI 2-sided [-1.89 to 1.35]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SOS-10 scores, t(326) = -1.28, d = 0.14; Test type: Superiority; p = 0.20, Mixed Models Analysis; Slope = -1.03, 95% CI 2-sided [-2.61 to 0.55]

19. Other Pre Specified Outcome: Change in Overall Self-Compassion Assessed Through the Self Compassion Scale (SCS)
Description: The Self Compassion Scale (SCS; Neff, 2003) is a 26-item measure that includes 6 subscales (including Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, and Over-Identification) and measures overall self-compassion. The possible range of scores is 1 to 5, with higher scores indicating higher self-compassion. The SCS has shown good internal consistency reliability as well as good test-retest reliability (Neff, 2003).
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 82 | 81
  Baseline | 2.66 (0.57) | 2.49 (0.56)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 2.97 (0.76) | 2.61 (0.64)
  3 month follow-up: number analyzed (Participants) | 47 | 52
  3 month follow-up | 3.01 (0.78) | 2.57 (0.68)
  6 month follow-up: number analyzed (Participants) | 40 | 39
  6 month follow-up | 3.13 (0.78) | 2.67 (0.61)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SCS scores, t(319) = 2.93, d = 0.33; Test type: Superiority; p = 0.004, Mixed Models Analysis; Slope = 0.26, 95% CI 2-sided [0.08 to 0.43]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for SCS scores, t(114) = 5.56, d = 1.04; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = 0.35, 95% CI 2-sided [0.23 to 0.48]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SCS scores, t(114) = 1.61, d = 0.30; Test type: Superiority; p = 0.11, Mixed Models Analysis; Slope = 0.10, 95% CI 2-sided [-0.02 to 0.22]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SCS scores, t(319) = 0.10, d = 0.10; Test type: Superiority; p = 0.92, Mixed Models Analysis; Slope = 0.007, 95% CI 2-sided [-0.13 to 0.15]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for SCS scores, t(319) = 0.31, d = 0.03; Test type: Superiority; p = 0.75, Mixed Models Analysis; Slope = 0.02, 95% CI 2-sided [-0.08 to 0.12]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SCS scores, t(319) = 0.18, d = 0.02; Test type: Superiority; p = 0.86, Mixed Models Analysis; Slope = 0.01, 95% CI 2-sided [-0.09 to 0.11]

20. Other Pre Specified Outcome: Change in State Anger Assessed Through the Dimensions of Anger Reactions (DAR)
Description: The Dimensions of Anger Reactions (DAR; Forbes et al., 2004) is a widely used measure of state anger. The measure consists of a 7-item inventory intended to capture anger disposition. Possible scores range from 0 to 56, with higher scores indicating higher state anger.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 85 | 81
  Baseline | 30.27 (12.90) | 32.32 (12.06)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 24.63 (13.96) | 29.07 (15.17)
  3 month follow-up: number analyzed (Participants) | 46 | 52
  3 month follow-up | 22.52 (14.53) | 28.96 (15.10)
  6 month follow-up: number analyzed (Participants) | 40 | 39
  6 month follow-up | 20.85 (14.28) | 28.51 (13.37)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for DAR scores, t(325) = -1.43, d = 0.16; Test type: Superiority; p = 0.15, Mixed Models Analysis; Slope = -2.56, 95% CI 2-sided [-6.10 to 0.97]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for DAR scores, t(116) = -4.07, d = 0.76; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -5.28, 95% CI 2-sided [-7.83 to -2.73]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for DAR scores, t(116) = -2.19, d = 0.41; Test type: Superiority; p = 0.03, Mixed Models Analysis; Slope = -2.71, 95% CI 2-sided [-5.16 to -0.28]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for DAR scores, t(325) = -0.97, d = 0.11; Test type: Superiority; p = 0.33, Mixed Models Analysis; Slope = -1.38, 95% CI 2-sided [-4.17 to 1.42]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for DAR scores, t(325) = -1.51, d = 0.17; Test type: Superiority; p = 0.13, Mixed Models Analysis; Slope = -1.54, 95% CI 2-sided [-3.54 to 0.46]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for DAR scores, t(325) = -0.17, d = 0.02; Test type: Superiority; p = 0.87, Mixed Models Analysis; Slope = -0.17, 95% CI 2-sided [-2.12 to 1.79]

21. Other Pre Specified Outcome: Change in Use of Psychologically Aggressive Behavior Assessed Through the Psychological Aggression Subscale of the Revised Conflict Tactics Scale (CTS2)
Description: The Psychological Aggression subscale of the Revised Conflict Tactics Scale (CTS2; Straus et al., 1996) was used to measure psychologically aggressive behavior. The subscales consists of 8 items, rated on a scale from 0 ("never") to 6 ("more than 20 times"), with higher scores indicating greater use of aggressive behaviors in the past month. To calculate the annual frequency score, values of 3 though 6 were transformed as follows: 3 = 4, 4 = 8, 5 = 15, 6 = 25. These values were then summed, with higher scores indicating greater frequency.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 85 | 82
  Baseline | 28.94 (31.45) | 26.41 (27.87)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 16.69 (22.19) | 19.47 (20.78)
  3 month follow-up: number analyzed (Participants) | 43 | 50
  3 month follow-up | 13.86 (20.40) | 17.84 (20.46)
  6 month follow-up: number analyzed (Participants) | 38 | 39
  6 month follow-up | 16.11 (23.64) | 17.77 (17.96)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CTS2 Psychological Aggression scores, t(319) = -2.03, d = 0.23; Test type: Superiority; p = 0.04, Mixed Models Analysis; Slope = -0.37, 95% CI 2-sided [-0.72 to -0.01]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for CTS2 Psychological Aggression scores, t(116)= -6.40, d = 1.19; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -0.83, 95% CI 2-sided [-1.09 to -0.58]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CTS2 Psychological Aggression scores, t(116) = -3.78, d = 0.70; Test type: Superiority; p = 0.002, Mixed Models Analysis; Slope = -0.47, 95% CI 2-sided [-0.71 to -0.22]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CTS2 Psychological Aggression scores, t(319) = -0.56, d = 0.06; Test type: Superiority; p = 0.58, Mixed Models Analysis; Slope = -0.08, 95% CI 2-sided [-0.37 to 0.21]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for CTS2 Psychological Aggression scores, t(319) = -0.96, d = 0.11; Test type: Superiority; p = 0.34, Mixed Models Analysis; Slope = -0.10, 95% CI 2-sided [-0.31 to 0.11]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CTS2 Psychological Aggression scores, t(319) = -0.19, d = 0.02; Test type: Superiority; p = 0.85, Mixed Models Analysis; Slope = -0.02, 95% CI 2-sided [-0.22 to 0.18]

22. Other Pre Specified Outcome: Change in Use of Physically Aggressive Behavior Assessed Through the Physical Assault Subscale on the Revised Conflict Tactics Scale (CTS2)
Description: The Physical Assault subscale of the Revised Conflict Tactics Scale (CTS2; Straus & Douglas, 2004; Straus et al., 1996) was used to measure occurrence of physically aggressive behavior. The subscale consists of 12 items, rated on a scale from 0 ("never") to 6 ("more than 20 times"), with higher scores indicating greater use of aggressive behaviors in the past month. To calculate the annual frequency score, values of 3 through 6 were transformed as follows: 3 = 4, 4 = 8, 5 = 15, 6 = 25. These values were then summed, with higher scores indicating greater frequency.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 85 | 82
  Baseline | 5.25 (30.27) | 0.96 (3.31)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 1.12 (3.33) | 1.64 (5.19)
  3 month follow up: number analyzed (Participants) | 43 | 50
  3 month follow up | 0.30 (1.28) | 4.10 (24.47)
  6 month follow up: number analyzed (Participants) | 38 | 39
  6 month follow up | 0.24 (0.91) | 1.69 (6.81)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CTS2 Physical Assault scores, t(319)= -1.82, d = 0.20; Test type: Superiority — We log-transformed CTS2 scores because they were heavily positively skewed in conjunction with zero-inflation; p = 0.07, Mixed Models Analysis; Slope = -0.23, 95% CI 2-sided [-0.48 to 0.02]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for CTS2 Physical Assault scores, t(116) = -1.39, d = 0.16; Test type: Superiority; p = 0.17, Mixed Models Analysis; Slope = -0.13, 95% CI 2-sided [-0.31 to -0.05]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CTS2 Physical Assault scores, t(116) = 1.18, d = 0.13; Test type: Superiority; p = 0.24, Mixed Models Analysis; Slope = 0.10, 95% CI 2-sided [-0.07 to 0.27]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CTS2 Physical Assault scores, t(319) = -0.37, d = 0.04; Test type: Superiority; p = 0.71, Mixed Models Analysis; Slope = 0.11, 95% CI 2-sided [-0.23 to 0.15]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for CTS2 Physical Assault scores, t(319) = -1.00, d = 0.11; Test type: Superiority; p = 0.32, Mixed Models Analysis; Slope = -0.07, 95% CI 2-sided [-0.21 to 0.07]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for CTS2 Physical Assault scores, t(319) = -0.51, d = 0.06; Test type: Superiority; p = 0.61, Mixed Models Analysis; Slope = -0.04, 95% CI 2-sided [-0.17 to 0.10]

23. Other Pre Specified Outcome: Change in Suicidality Across Assessed Through the Depressive Symptoms Index - Suicidality Subscale (DSI-SS)
Description: The Depressive Symptoms Index - Suicidality Subscale (DSI-SS; Metalsky & Joiner, 1997) is a 4-item scale that focuses on ideation, plans, perceived control over ideation, and impulses for suicide. A review of measures of suicidal ideation and behaviors found that the DSI-SS had excellent internal consistency and concurrent validity (Batterham et al., 2014). Possible scores range from 0 to 12, with higher scores indicating greater severity of suicidal ideation.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after posttreatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 81 | 82
  Baseline | 1.14 (1.62) | 0.93 (1.65)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 1.00 (1.63) | 0.85 (1.55)
  3 month follow-up: number analyzed (Participants) | 47 | 51
  3 month follow-up | 0.91 (1.61) | 0.94 (1.58)
  6 month follow-up: number analyzed (Participants) | 40 | 39
  6 month follow-up | 1.15 (1.72) | 1.05 (1.62)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for DSI-SS scores, t(318) = -0.33, d = 0.04; Test type: Superiority; p = 0.74, Mixed Models Analysis; Slope = -0.07, 95% CI 2-sided [-0.50 to 0.36]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for DSI-SS scores, t(114) = -0.77, d = 0.14; Test type: Superiority; p = 0.44, Mixed Models Analysis; Slope = -0.12, 95% CI 2-sided [-0.43 to 0.19]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for DSI-SS scores, t(114) = -0.34, d = 0.06; Test type: Superiority; p = 0.74, Mixed Models Analysis; Slope = -0.06, 95% CI 2-sided [-0.35 to 0.24]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for DSI-SS scores, t(114) = -0.57, d = 0.11; Test type: Superiority; p = 0.57, Mixed Models Analysis; Slope = -0.10, 95% CI 2-sided [-0.45 to 0.25]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for DSI-SS scores, t(114) = -0.23, d = 0.04; Test type: Superiority; p = 0.82, Mixed Models Analysis; Slope = -0.03, 95% CI 2-sided [-0.28 to 0.22]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for DSI-SS scores, t(114) = 0.58, d = 0.11; Test type: Superiority; p = 0.57, Mixed Models Analysis; Slope = 0.07, 95% CI 2-sided [-0.17 to 0.31]

24. Other Pre Specified Outcome: Change in Alcohol Consumption Assessed Through the Quick Drinking Screen (QDS)
Description: Alcohol abuse was evaluated with the Quick Drinking Screen (QDS; Sobell et al., 2003), a 4-item probe of frequency and quantity of alcohol consumption in the last month. The QDS has very good psychometric characteristics (Sobell et al., 2003). The outcome for this measure used in this study was average drinks per week, calculated by using items 1 and 2 from the screen.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Estimated drinks per week
Groups:
- Present Centered Therapy: Participants randomized to the PCT arm received 12 sessions of therapy focused on improving day-to-day functioning (with no focus on trauma or re-visiting past experiences). PCT is a manualized evidenced-based PTSD treatment used in several large-scale PTSD trials that focuses on improving functioning. It incorporates the essential therapeutic elements common to different types of psychotherapies, including supportive empathic listening and unconditional positive regard. The therapist plays an active role but does not impart any systematic training. The focus is to create an understanding of how the symptoms of PTSD are related to day-to-day difficulties and to help patients develop new, more adaptive functional responses to these stressors with a problem-focused and problem- solving approach. In prior trials, PCT showed equivalent change to active therapies at the last follow-up. The VA offers PCT as an evidence-based therapy for PTSD.
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Estimated drinks per week
  Baseline: number analyzed (Participants) | 85 | 82
  Baseline | 1.92 (3.17) | 1.97 (2.81)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 0.84 (1.58) | 2.16 (3.55)
  3 month follow-up: number analyzed (Participants) | 43 | 50
  3 month follow-up | 1.27 (2.28) | 2.37 (4.34)
  6 month follow-up: number analyzed (Participants) | 37 | 39
  6 month follow-up | 0.84 (1.87) | 2.55 (4.81)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for QDS scores, t(316) = -1.42, d = 0.16; Test type: Superiority; p = 0.16, Mixed Models Analysis; Slope = -1.10, 95% CI 2-sided [-2.63 to 0.43]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for QDS scores, t(114)= -1.35, d = 0.25; Test type: Superiority; p = 0.18, Mixed Models Analysis; Slope = -0.76, 95% CI 2-sided [-1.87 to 0.35]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for QDS scores, t(114) = 0.63, d = 0.12; Test type: Superiority; p = 0.53, Mixed Models Analysis; Slope = 0.34, 95% CI 2-sided [-0.71 to 1.39]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for QDS scores, t(316) = -0.89, d = 0.12; Test type: Superiority; p = .37, Mixed Models Analysis; Slope = -0.60, 95% CI 2-sided [-1.93 to 0.73]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for QDS scores, t(114) = -0.08, d = 0.02; Test type: Superiority; p = 0.94, Mixed Models Analysis; Slope = -0.04, 95% CI 2-sided [-1.00 to 0.92]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for QDS scores, t(114) = 1.21, d = 0.23; Test type: Superiority; p = 0.23, Mixed Models Analysis; Slope = 0.57, 95% CI 2-sided [-0.35 to 1.48]

25. Other Pre Specified Outcome: Change in Social Connectedness Assessed Through the Social Connectedness Scale (SCS)
Description: The Social Connectedness Scale (SCS; Lee and Robbins, 1995) was used to assess interpersonal closeness. The SCS is an 8-item scale that focuses on individual experiences in a social world (i.e., with peers, friends, and society) and the degree of difficulty in maintaining a sense of closeness. Possible scores range from 8 to 42, with higher scores indicating more social connection.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 85 | 82
  Baseline | 23.89 (9.69) | 23.56 (8.22)
  Post treatment: number analyzed (Participants) | 48 | 59
  Post treatment | 28.08 (11.75) | 24.78 (9.16)
  3 month follow-up: number analyzed (Participants) | 43 | 50
  3 month follow-up | 29.56 (12.11) | 26.41 (10.83)
  6 month follow-up: number analyzed (Participants) | 38 | 39
  6 month follow-up | 29.83 (12.17) | 27.21 (9.10)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SCS scores, t(316) = 2.49, d = 0.28; Test type: Superiority; p = 0.01, Mixed Models Analysis; Slope = 3.98, 95% CI 2-sided [0.83 to 7.13]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for SCS scores, t(114) = 4.16, d = 0.78; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = 4.84, 95% CI 2-sided [2.55 to 7.13]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SCS scores, t(114) = 0.78, d = 0.15; Test type: Superiority; p = 0.44, Mixed Models Analysis; Slope = 0.85, 95% CI 2-sided [-1.31 to 3.02]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SCS scores, t(316) = 0.17, d = 0.02; Test type: Superiority; p = 0.88, Mixed Models Analysis; Slope = 0.21, 95% CI 2-sided [-2.32 to 2.75]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for SCS scores, t(316) = 0.60, d = 0.07; Test type: Superiority; p = 0.55, Mixed Models Analysis; Slope = 0.55, 95% CI 2-sided [-1.27 to 2.37]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SCS scores, t(316) = 0.38, d = 0.04; Test type: Superiority; p = 0.70, Mixed Models Analysis; Slope = 0.38, 95% CI 2-sided [-1.42 to 2.10]

26. Other Pre Specified Outcome: Change in Compassion for Humanity Assessed Through The Santa Clara Brief Compassion Scale (SCBSC)
Description: The Santa Clara Brief Compassion Scale (SCBSC; Hwang, et al., 2008) is a 5-item short form of the Compassionate Love Scale for Humanity (CLS). Possible scores range from 1 to 7, with higher scores indicating more compassion for humanity.
Time Frame: Assessments occurred at baseline, post treatment, and approximately 3 and 6 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a scale
  Baseline: number analyzed (Participants) | 85 | 82
  Baseline | 4.84 (1.76) | 5.00 (1.64)
  Post treatment: number analyzed (Participants) | 49 | 59
  Post treatment | 4.93 (1.65) | 5.02 (1.63)
  3 month follow-up: number analyzed (Participants) | 43 | 50
  3 month follow-up | 5.12 (1.56) | 4.82 (1.77)
  6 month follow-up: number analyzed (Participants) | 38 | 39
  6 month follow-up | 4.97 (1.73) | 4.85 (1.54)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SCBSC scores, t(318) = -0.25, d = 0.03; Test type: Superiority; p = 0.80, Mixed Models Analysis; Slope = -0.04, 95% CI 2-sided [-0.32 to 0.25]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for SCBSC scores, t(115) = 0.57, d = 0.11; Test type: Superiority; p = 0.57, Mixed Models Analysis; Slope = 0.04, 95% CI 2-sided [-0.09 to 0.16]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SCBSC scores, t(115) = -0.23, d = 0.04; Test type: Superiority; p = 0.82, Mixed Models Analysis; Slope = -0.01, 95% CI 2-sided [-0.14 to 0.11]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for SCBSC scores, t(320) = 0.57, d = 0.06; Test type: Superiority; p = 0.57, Mixed Models Analysis; Slope = 0.05, 95% CI 2-sided [-0.13 to 0.23]

27. Post Hoc Outcome: Change in Valued/Mindful Living Assessed Through The Valued Living Questionnaire (VLQ)
Description: The Valued Living Questionnaire (VLQ; Wilson et al., 2010) value and engagement in 10 domains of living. Respondents rate how important each domain is from 1 ("not at all important") to 10 ("extremely important"; Importance subscale) and their engagement in each domain, on a scale from 1 ("not at all consistent with my value") to 10 ("completely consistent with my value"; Consistency subscale). Importance and Consistency scores are multiplied for each domain, added across domains, and then divided by 10 such that possible scores range from 10-100. Higher scores indicate greater valued living.
Time Frame: Assessments occurred at baseline, the sixth treatment session, post treatment, and approximately 3 months after post treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a composite scale
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
Number analyzed (Participants) | 89 | 85
Score on a composite scale
  Baseline: number analyzed (Participants) | 79 | 81
  Baseline | 37.39 (19.42) | 40.72 (16.89)
  Session 6: number analyzed (Participants) | 57 | 57
  Session 6 | 42.42 (18.02) | 40.51 (16.31)
  Post treatment: number analyzed (Participants) | 50 | 56
  Post treatment | 47.32 (19.80) | 43.81 (18.96)
  3 month follow up: number analyzed (Participants) | 47 | 52
  3 month follow up | 46.24 (20.72) | 44.10 (20.33)
  6 month follow up: number analyzed (Participants) | 40 | 38
  6 month follow up | 44.42 (19.40) | 45.29 (21.33)
Statistical Analysis 1: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for VLQ scores, t(408) = 3.16, d = 0.32; Test type: Superiority; p = 0.002, Mixed Models Analysis; Slope = 3.91, 95% CI 2-sided [1.48 to 6.35]
Statistical Analysis 2: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for VLQ scores, t(121) = 4.66, d = 0.85; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = 4.16, 95% CI 2-sided [2.41 to 5.92]
Statistical Analysis 3: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for VLQ scores, t(121) = 0.63, d = 0.11; Test type: Superiority; p = 0.78, Mixed Models Analysis; Slope = 0.25, 95% CI 2-sided [-1.44 to 1.94]
Statistical Analysis 4: Comparison: Adaptive Disclosure for Moral Injury and Loss vs Present Centered Therapy; In a mixed model analysis of intent-to-treat data for VLQ scores, t(408) = -0.34, d = 0.01; Test type: Superiority; p = 0.73, Mixed Models Analysis; Slope = -0.05, 95% CI 2-sided [-0.34 to 0.24]
Statistical Analysis 5: Comparison: Adaptive Disclosure for Moral Injury and Loss; In a mixed model analysis of intent-to-treat data for VLQ scores, t(408) = 0.56, d = 0.06; Test type: Superiority; p = 0.58, Mixed Models Analysis; Slope = 0.06, 95% CI 2-sided [-0.15 to 0.27]
Statistical Analysis 6: Comparison: Present Centered Therapy; In a mixed model analysis of intent-to-treat data for VLQ scores, t(408) = 1.07, d = 0.11; Test type: Superiority; p = 0.28, Mixed Models Analysis; Slope = 0.11, 95% CI 2-sided [-0.10 to 0.31]

ADVERSE EVENTS:
Time Frame: Adverse event data for a given participant were collected for the entire period that the participant was involved in the study. Adverse events were monitored for from the time consent was collected through the duration of the clinical intervention, which, for participants who completed the entire study, was approximately 9 months. For all participants combined, data were collected for approximately 4 years (January 2018-January 2022).
Description: All adverse events, both serious and non serious, regardless of relationship to the study intervention, were recorded on the VA Boston IRB adverse event log. Adverse event data were collected from the time the informed consent form is signed through the duration of the clinical investigation. Standard medical terminology was used when recording Adverse events.
Arm/Group | Adaptive Disclosure for Moral Injury and Loss | Present Centered Therapy
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/85
Serious Adverse Events (participants affected / at risk) | 1/89 | 2/85
Other Adverse Events (participants affected / at risk) | 7/89 | 10/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adaptive Disclosure for Moral Injury and Loss (N=89) | Present Centered Therapy (N=85)
Hospitalization due to hypertension/elevated heart rate (Cardiac disorders) | 0 (0) | 1 (1) — Hospitalization due to hypertension/elevated heart rate. Hx of high BP & other physical health concerns noted in chart. Issue ongoing as of 9/30/2019
Pt relapsed on alcohol and self-admitted to a 30-day rehabilitation program (Psychiatric disorders) | 0 (0) | 1 (1)
Right small toe was amputated due to an infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adaptive Disclosure for Moral Injury and Loss (N=89) | Present Centered Therapy (N=85)
Increase in psychiatric symptoms (Psychiatric disorders) | 7 (10) | 10 (11)

LIMITATIONS AND CAVEATS:
Therapists delivered both therapies; Did not measure moral injury or prolonged grief as outcomes; Approximately half of participants were not evaluated at the 6-month follow-up interval; Use of retrospective paper and pencil measures of functioning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT03056157/Prot_SAP_ICF_000.pdf